CLINICAL TRIAL: NCT01262872
Title: Impact of GSK Biologicals' 2189242A Vaccine on Nasopharyngeal Carriage, Safety and Immunogenicity When Co-administered With Routine EPI Vaccines in Infants Following Safety Assessment in Children Aged 2-4 Years in The Gambia
Brief Title: Impact of GSK Biologicals' 2189242A Vaccine on Nasopharyngeal Carriage, Safety & Immunogenicity in Children & Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PATH (Other); Department of State for Health and Social Welfare, The Gambia (Other Government); Medical Research Council Unit, The Gambia (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 114174; 2012-002727-15 (EudraCT Number)
Record Dates: First submitted 2010-12-02; First posted 2010-12-17 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Infections, Streptococcal
Keywords: Haemophilus influenzae; Streptococcus pneumoniae; The Gambia; immunogenicity; nasopharyngeal carriage; infants; safety; Pneumococcal vaccine; children
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections | interventions — PHiD-CV vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- 10PP-HD 1d Group (Experimental): This group consisted in children aged 2-4 years at vaccination enrolled as part of the Cohort 1/Step 1 of the study who received a single dose of the GSK 2189242A (or 10PP) vaccine in its high-dose (HD) formulation at Day 0. The 10PP vaccine was administered intramuscularly in the non-dominant deltoid.
  Interventions: Biological: Pneumococcal vaccine GSK 2189242A (HD formulation 2)
- Prevnar13 1d Group (Active Comparator): This group consisted in children aged 2-4 years at vaccination enrolled as part of the Cohort 1/Step 1 of the study who received a single dose of Prevnar 13™ at Day 0. Prevnar 13™ was administered intramuscularly in the non-dominant deltoid.
  Interventions: Biological: Prevnar13™
- 10PP-LD 3+0d Group (Experimental): This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received 3 doses of the GSK 2189242A (or 10PP) vaccine in its low-dose (LD) formulation and EPI vaccines according to a 3+0 Schedule. That is, subjects received 3 doses of the 10PP vaccine, LD formulation, co-administered with Tritanrix™-HepB/Hib and Polio Sabin™ at 2-3-4 months of age (Day 0, Month 1 and Month 2), followed by one dose of each of the M-Vac™, Stamaril™ and Polio Sabin™ vaccines administered at approximately 9 months of age. The 10PP vaccine was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
  Interventions: Biological: Pneumococcal vaccine GSK 2189242A (LD formulation 1); Biological: Tritanrix™-HepB/Hib; Biological: Polio Sabin™; Biological: M-Vac™; Biological: Stamaril™
- 10PP-HD 3+0d Group (Experimental): This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received 3 doses of the GSK 2189242A (or 10PP) vaccine in its high-dose (HD) formulation and EPI vaccines according to a 3+0 Schedule. That is, subjects received 3 doses of the 10PP vaccine, HD formulation, co-administered with the Tritanrix™-HepB/Hib and Polio Sabin™ at 2-3-4 months of age (Day 0, Month 1 and Month 2), followed by one dose of each of the M-Vac™, Stamaril™ and Polio Sabin™ vaccines administered at approximately 9 months of age. The 10PP vaccine was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
  Interventions: Biological: Pneumococcal vaccine GSK 2189242A (HD formulation 2); Biological: Tritanrix™-HepB/Hib; Biological: Polio Sabin™; Biological: M-Vac™; Biological: Stamaril™
- Synflorix 3+0d Group (Active Comparator): This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received 3 doses of Synflorix™ and EPI vaccines according to a 3+0 Schedule. That is, subjects received 3 doses of the Synflorix™, co-administered with Tritanrix™-HepB/Hib and Polio Sabin™ at 2-3-4 months of age (Day 0, Month 1 and Month 2), followed by one dose of each of the M-Vac™, Stamaril™ and Polio Sabin™ vaccines administered at approximately 9 months of age. Synflorix™ was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
  Interventions: Biological: Synflorix™; Biological: Tritanrix™-HepB/Hib; Biological: Polio Sabin™; Biological: M-Vac™; Biological: Stamaril™
- Prevnar13 3+0d Group (Active Comparator): This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received 3 doses of Prevnar 13™ and EPI vaccines according to a 3+0 Schedule. That is, subjects received 3 doses of Prevnar 13™, co-administered with Tritanrix™-HepB/Hib and Polio Sabin™ at 2-3-4 months of age (Day 0, Month 1 and Month 2), followed by one dose of each of the M-Vac™, Stamaril™ and Polio Sabin™ vaccines administered at approximately 9 months of age. Prevnar 13™ was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
  Interventions: Biological: Prevnar13™; Biological: Tritanrix™-HepB/Hib; Biological: Polio Sabin™; Biological: M-Vac™; Biological: Stamaril™
- 10PP-HD 2+1d Group (Experimental): This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received the GSK 2189242A (or 10PP) vaccine, in its high-dose (HD) formulation, and EPI vaccines according to a 2+1 Schedule. That is, subjects received 2 doses of the 10PP vaccine, HD formulation co-administered with Tritanrix™-Hep B/Hib and Polio Sabin™ at 2-4 months of age (at Day 0 and Month 2), followed by a third dose of the same formulation co-administered with M-Vac™, Stamaril™ and Polio Sabin™ at approximately 9 months of age.. The 2nd doses of Tritanrix™-Hep B/Hib and Polio Sabin™ in EPI vaccines were administered without any pneumococcal vaccine at 3 months of age. The 10PP vaccine was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
  Interventions: Biological: Pneumococcal vaccine GSK 2189242A (HD formulation 2); Biological: Tritanrix™-HepB/Hib; Biological: Polio Sabin™; Biological: M-Vac™; Biological: Stamaril™
- Synflorix 2+1d Group (Active Comparator): This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received Synflorix™ and EPI vaccines according to a 2+1 Schedule. That is, subjects received 2 doses of the Synflorix™ co-administered with Tritanrix™-Hep B/Hib and Polio Sabin™ at 2-4 months of age (at Day 0 and Month 2), followed by a third dose of Synflorix™ co-administered with M-Vac™, Stamaril™ and Polio Sabin™ at approximately 9 months of age. The 2nd doses of Tritanrix™-Hep B/Hib and Polio Sabin™ in EPI vaccines were administered without any pneumococcal vaccine at 3 months of age. Synflorix™ was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
  Interventions: Biological: Synflorix™; Biological: Tritanrix™-HepB/Hib; Biological: Polio Sabin™; Biological: M-Vac™; Biological: Stamaril™

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK 2189242A (LD formulation 1) — Intramuscular injection
  Other Names: 10PP; LD Formulation
  Arms: 10PP-LD 3+0d Group
Biological: Pneumococcal vaccine GSK 2189242A (HD formulation 2) — Intramuscular injection
  Other Names: 10PP; HD Formulation
  Arms: 10PP-HD 1d Group; 10PP-HD 2+1d Group; 10PP-HD 3+0d Group
Biological: Synflorix™ — Intramuscular injection
  Arms: Synflorix 2+1d Group; Synflorix 3+0d Group
Biological: Prevnar13™ — Intramuscular injection
  Arms: Prevnar13 1d Group; Prevnar13 3+0d Group
Biological: Tritanrix™-HepB/Hib — Intramuscular injection
  Arms: 10PP-HD 2+1d Group; 10PP-HD 3+0d Group; 10PP-LD 3+0d Group; Prevnar13 3+0d Group; Synflorix 2+1d Group; Synflorix 3+0d Group
Biological: Polio Sabin™ — Orally
  Arms: 10PP-HD 2+1d Group; 10PP-HD 3+0d Group; 10PP-LD 3+0d Group; Prevnar13 3+0d Group; Synflorix 2+1d Group; Synflorix 3+0d Group
Biological: M-Vac™ — Intramuscular injection
  Arms: 10PP-HD 2+1d Group; 10PP-HD 3+0d Group; 10PP-LD 3+0d Group; Prevnar13 3+0d Group; Synflorix 2+1d Group; Synflorix 3+0d Group
Biological: Stamaril™ — Intramuscular injection
  Arms: 10PP-HD 2+1d Group; 10PP-HD 3+0d Group; 10PP-LD 3+0d Group; Prevnar13 3+0d Group; Synflorix 2+1d Group; Synflorix 3+0d Group

SUMMARY:
This study will assess the impact on nasopharyngeal carriage, safety and immunogenicity of GSK Biologicals' pneumococcal vaccine 2189242A given as a 3-dose vaccination course and co-administered with other routine paediatric vaccines in infants in The Gambia. Two formulations containing different doses of pneumococcal antigen and two different schedules will be tested in infants.

DETAILED DESCRIPTION:
There will be two cohorts in the study: Cohort 1 (children aged 2-4 years) and Cohort 2 (infants aged 8-10 weeks), and two steps in the study, Step 1 and Step 2. Step 1 will consist in a safety evaluation of the GSK Biologicals' pneumococcal vaccine 2189242A (GSK 2189242A or 10PP vaccine). Before evaluating the two formulations of the 10PP vaccine in infants (Cohort 2), safety and reactogenicity of the highest dose formulation of this vaccine will be evaluated in children (Cohort 1). Prevnar 13™ will be used as a control. In the second step of the study, Step 2, two investigational formulations of the 10PP vaccine will be tested in infants (Cohort 2) as regards immunogenicity, reactogenicity and safety. Both formulations of the 10PP vaccine will be evaluated according to the Expanded Programme on Immunization (EPI) schedule i.e. a 2, 3, 4 months vaccination schedule, using licensed Synflorix™ and Prevnar 13™ vaccines as comparators. The higher dose (HD) formulation of the 10PP vaccine will be also evaluated according to the 2, 4, 9 months vaccination schedule using licensed Synflorix™ vaccine as comparator. The study in infants will also assess the immune responses to routine vaccines when co-administered with the candidate pneumococcal vaccine, using licensed Synflorix™ and Prevnar 13™ vaccines as comparators.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for subjects in Cohort 1 (children) and Cohort 2 (infants):

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol
* Male or female between, and including,

  * 2 to 4 years of age at the time of the first vaccination for subjects in Cohort 1 (children).
  * 8 to 10 weeks (56-76 days) of age at the time of the first vaccination for subjects in Cohort 2 (infants).
* Signed or thumb-printed informed consent obtained from the parents/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Permanent residence in the study area and no intention of leaving during the study period.

Additional inclusion criteria for subjects in Cohort 1:

• Previously completed three-dose primary course of diphtheria-tetanus-pertussis (DTP) vaccination.

Exclusion Criteria:

Exclusion criteria for subjects in Cohort 1 (children) and Cohort 2 (infants):

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the study period starting from 30 days before each dose and ending 30 days after each dose of vaccine(s), with the exception of licensed flu vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Previous vaccination against S. pneumoniae.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Malnutrition
* A family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or any chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/ or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Contraindications to any co-administered vaccine.
* Any medical condition that would contraindicate the initiation of routine immunization outside a clinical trial context.

Additional exclusion criteria for subjects in Cohort 1:

• Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b with the exception of vaccines where the first dose should be given within the first two weeks of life according to the national recommendations (for example Bacillus Calmette-Guérin [BCG] and hepatitis B vaccination).

Ages: 56 Days to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1320 (Actual)
Dates: Start 2011-02-09 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Odutola A, Antonio M, Owolabi O, Bojang A, Foster-Nyarko E, Donkor S, Adetifa I, Taylor S, Bottomley C, Greenwood B, Ota M. Comparison of the prevalence of common bacterial pathogens in the oropharynx and nasopharynx of gambian infants. PLoS One. 2013 Sep 23;8(9):e75558. doi: 10.1371/journal.pone.0075558. eCollection 2013. PMID 24086570
- [Background] Odutola A, Ota MO, Ogundare EO, Antonio M, Owiafe P, Worwui A, Greenwood B, Alderson M, Traskine M, Verlant V, Dobbelaere K, Borys D. Reactogenicity, safety and immunogenicity of a protein-based pneumococcal vaccine in Gambian children aged 2-4 years: A phase II randomized study. Hum Vaccin Immunother. 2016;12(2):393-402. doi: 10.1080/21645515.2015.1111496. PMID 26618243
- [Background] Odutola A, Ota MOC, Antonio M, Ogundare EO, Saidu Y, Foster-Nyarko E, Owiafe PK, Ceesay F, Worwui A, Idoko OT, Owolabi O, Bojang A, Jarju S, Drammeh I, Kampmann B, Greenwood BM, Alderson M, Traskine M, Devos N, Schoonbroodt S, Swinnen K, Verlant V, Dobbelaere K, Borys D. Efficacy of a novel, protein-based pneumococcal vaccine against nasopharyngeal carriage of Streptococcus pneumoniae in infants: A phase 2, randomized, controlled, observer-blind study. Vaccine. 2017 May 2;35(19):2531-2542. doi: 10.1016/j.vaccine.2017.03.071. Epub 2017 Apr 4. PMID 28389097
- [Background] Odutola A, Ota MOC, Antonio M, Ogundare EO, Saidu Y, Owiafe PK, Worwui A, Idoko OT, Owolabi O, Kampmann B, Greenwood BM, Alderson M, Traskine M, Swinnen K, Verlant V, Dobbelaere K, Borys D. Immunogenicity of pneumococcal conjugate vaccine formulations containing pneumococcal proteins, and immunogenicity and reactogenicity of co-administered routine vaccines - A phase II, randomised, observer-blind study in Gambian infants. Vaccine. 2019 May 1;37(19):2586-2599. doi: 10.1016/j.vaccine.2019.03.033. Epub 2019 Apr 8. PMID 30975570
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114174 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114174 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114174 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114174 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114174 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114174 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 subjects participated in Step 1 (duration of about 6 months). Cohort 2 subjects participated in Step 2 (duration of about 10 months). Enrolment for Step 2 was conditional upon successful results of a post-vaccination safety evaluation of all children enrolled in Cohort 1 by an Independent Data Monitoring Committee.
Pre-assignment Details: Description of any significant events and approaches for the overall study following participant enrollment, but prior to group assignment.
Period: Step 1
Arm/Group | 10PP-HD 1d Group | Prevnar13 1d Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Started | 60 | 60 | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.)
Completed | 60 | 60 | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 2
Arm/Group | 10PP-HD 1d Group | Prevnar13 1d Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Started | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 200 | 200 | 200 | 200 | 200 | 200
Completed | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 0 (The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone.) | 191 | 190 | 195 | 191 | 191 | 194
Not Completed | 0 | 0 | 9 | 10 | 5 | 9 | 9 | 6
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 6 | 3 | 1 | 2 | 1
Not completed — Migrated/moved from study area | 0 | 0 | 4 | 3 | 2 | 6 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10PP-HD 1d Group | Prevnar13 1d Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group | Total
Number analyzed (Participants) | 60 | 60 | 200 | 200 | 200 | 200 | 200 | 200 | 1320
Age, Continuous [Mean (Standard Deviation); unit: Years] | 2.8 (0.40) | 2.9 (0.36) | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | 2.9 (0.38)
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA (NA) — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | 8.5 (0.64) | 8.4 (0.61) | 8.4 (0.63) | 8.5 (0.69) | 8.5 (0.70) | 8.5 (0.70) | 8.5 (0.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 26 | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 19 | 34 | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | 105 | 98 | 103 | 103 | 103 | 97 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | 95 | 102 | 97 | 97 | 97 | 103 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage | 60 | 60 | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | NA — The 2 first groups included subjects for Step 1 alone. The 6 other groups were part of Step 2 alone. | 200 | 200 | 200 | 200 | 200 | 200 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms and Grade 3 Solicited Local Symptoms With Relationship to Vaccination - For Step 1/Cohort 1 Subjects
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm). All solicited local symptoms were systematically considered by the investigators as causally related to vaccination. Primary results correspond to results for occurrences of Grade 3 symptoms. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: Within the 4-day (Days 0-3) period post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 1d Group | Prevnar13 1d Group
Number analyzed (Participants) | 60 | 60
Participants
  Any Pain | 0 | 0
  Grade 3 Pain | 0 | 0
  Any Redness | 0 | 0
  Grade 3 Redness | 0 | 0
  Any Swelling | 1 | 0
  Grade 3 Swelling | 1 | 0

2. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms With and Without Relationship to Vaccination - For Step 1/Cohort 1 Subjects
Description: Assessed solicited general symptoms were Drowsiness, Fever (axillary temperature higher than [≥] 37.5 degrees Celsius [°C]), Irritability/Fussiness and Loss of appetite. Any = Occurrence of the specified solicited general symptom, regardless of intensity and relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigator as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Fever = Axillary temperature higher than (>) 39.5°C. Grade 3 Irritability/fussiness = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Primary results correspond to results for occurrences of Grade 3 symptoms assessed as related to vaccination. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: Within the 4-day (Days 0-3) period post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 1d Group | Prevnar13 1d Group
Number analyzed (Participants) | 60 | 60
Participants
  Any Drowsiness | 0 | 0
  Grade 3 Drowsiness | 0 | 0
  Related Drowsiness | 0 | 0
  Grade 3 & Related Drowsiness | 0 | 0
  Any Fever | 4 | 2
  Grade 3 Fever | 0 | 0
  Related Fever | 1 | 1
  Grade 3 & Related Fever | 0 | 0
  Any Irritability/Fussiness | 0 | 0
  Grade 3 Irritability/Fussiness | 0 | 0
  Related Irritability/Fussiness | 0 | 0
  Grade 3 & Related Irritability/Fussiness | 0 | 0
  Any Loss of appetite | 1 | 0
  Grade 3 Loss of appetite | 0 | 0
  Related Loss of appetite | 0 | 0
  Grade 3 & Related Loss of appetite | 0 | 0

3. Primary Outcome: Number of Subjects With Any and Grade 3 Unsolicited Adverse Events (AEs) With and Without Relationship to Vaccination - In Step 1/Cohort 1 Subjects
Description: An unsolicited AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. Any = Occurrence of AE, regardless of intensity or relationship to vaccination. Grade 3 = Occurrence of AE which prevented normal activities. Related = Occurrence of AE assessed by the investigator as causally related to vaccination. Primary results correspond to results for occurrences of Grade 3 unsolicited AE(s) assessed as related to vaccination. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: Within the 31-day (Days 0-30) period post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 1d Group | Prevnar13 1d Group
Number analyzed (Participants) | 60 | 60
Participants
  Any unsolicited AE(s) | 13 | 7
  Grade 3 unsolicited AE(s) | 0 | 0
  Related unsolicited AE(s) | 0 | 0
  Grade 3 and related unsolicited AE(s) | 0 | 0

4. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) and With SAE(s) With Relationship to Vaccination - In Step 1/Cohort 1 Subjects
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity. These should also be considered serious: invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation. Any = Occurrence of an SAE, regardless of relationship to vaccination. Related = Occurrence of an SAE assessed by the investigator as causally related to vaccination. Primary results correspond to results for occurrences of SAE(s) assessed as related to vaccination. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: From Day 0 to Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Prevnar 13 1d Group: This group consisted in children aged 2-4 years at vaccination enrolled as part of the Cohort 1/Step 1 of the study who received a single dose of Prevnar 13™ at Day 0. Prevnar 13™ was administered intramuscularly in the non-dominant deltoid.
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group
Number analyzed (Participants) | 60 | 60
Participants
  Any SAE(s) | 0 | 0
  SAE(s) related to vaccination | 0 | 0

5. Primary Outcome: Number of Subjects With Non-vaccine Serotypes of Streptococcus Pneumoniae (S. pn.) in the Nasopharynx - For Cohort 2/Step 2, Subjects Receiving the 3+0 Schedule
Description: Any serotype belonging to the same serogroup as the serotypes of the pneumococcal vaccine administered (10PP vaccine or Synflorix™), but different from 10 vaccine pneumococcal serotypes, was considered for this analysis of carriage. Serotypes were identified through cultures and serotyping of the isolates.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196
Participants
  1 Mth post dose 3 | 154 | 137 | 145
  5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 194
  5 Mth post dose 3 | 148 | 149 | 159
  8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194
  8 Mth post dose 3 | 151 | 154 | 159
Statistical Analysis 1: Comparison: 10PP-LD 3+0d Group vs Synflorix 3+0d Group; VE-10PP-LD 3+0d vs Synflorix 3+0d - 1M post-Dose 3. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, one month (M) post-dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — Vaccine efficacy (VE) estimated as [(1-Relative Risk (i.e. investigational vaccine over control vaccine))*100] with 95% CI was calculated. Denominator considered for deriving VE at a considered time point was the number of subjects with swabs cultured at this time point. Power using 2 independent proportions, 1:1 randomization ratio, 1-sided test to detect group difference, 1-sided alpha=2.5%; VE = -7.9, 95% CI 2-sided [-36.3 to 14.6]
Statistical Analysis 2: Comparison: 10PP-LD 3+0d Group vs Synflorix 3+0d Group; VE-10PP-LD 3+0d vs Synflorix 3+0d - 5M post-Dose 3. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, five months (M) post-dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE = 6.4, 95% CI 2-sided [-17.8 to 25.7]
Statistical Analysis 3: Comparison: 10PP-LD 3+0d Group vs Synflorix 3+0d Group; VE-10PP-LD 3+0d vs Synflorix 3+0d - 8M post-Dose 3. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, eight months (M) post-dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE = 2.5, 95% CI 2-sided [-22.6 to 22.5]
Statistical Analysis 4: Comparison: 10PP-HD 3+0d Group vs Synflorix 3+0d Group; VE-10PP-HD 3+0d vs Synflorix 3+0d - 1M post-Dose 3. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, one month (M) post-dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE = 4.5, 95% CI 2-sided [-21.4 to 25.0]
Statistical Analysis 5: Comparison: 10PP-HD 3+0d Group vs Synflorix 3+0d Group; VE-10PP-HD 3+0d vs Synflorix 3+0d - 5M post-Dose 3. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, five months (M) post-dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE = 5.3, 95% CI 2-sided [-19.2 to 24.8]
Statistical Analysis 6: Comparison: 10PP-HD 3+0d Group vs Synflorix 3+0d Group; VE-10PP-HD 3+0d vs Synflorix 3+0d - 8M post-Dose 3. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, eight months (M) post-dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE = 0.6, 95% CI 2-sided [-24.9 to 20.9]

6. Primary Outcome: Number of Subjects With Non-vaccine Serotypes of Streptococcus Pneumoniae (S. pn.) in the Nasopharynx - For Cohort 2/Step 2, Subjects Receiving the 2+1 Schedule
Description: Any serotype belonging to the same serogroup as the serotypes of the pneumococcal vaccine administered (10PP vaccine or Synflorix™), but different from 10 vaccine pneumococcal serotypes, was considered for this analysis of carriage. Serotypes were identified through cultures and serotyping of isolates.
Time Frame: At 1 and 5 months (Mth) post-Dose 2, and at 3 months post-Dose 3 of the pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  1 Mth post dose 2 | 142 | 152
  5 Mth post dose 2: number analyzed (Participants) | 189 | 194
  5 Mth post dose 2 | 146 | 160
  3 Mth post dose 3: number analyzed (Participants) | 190 | 193
  3 Mth post dose 3 | 165 | 162
Statistical Analysis 1: Comparison: 10PP-HD 2+1d Group vs Synflorix 2+1d Group; VE-10PP-HD 2+1d vs Synflorix 2+1d - 1M post-Dose 2. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, one month (M) post-dose 2 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE (see above) = 6.6, 95% CI 2-sided [-18.2 to 26.2]
Statistical Analysis 2: Comparison: 10PP-HD 2+1d Group vs Synflorix 2+1d Group; VE-10PP-HD 2+1d vs Synflorix 2+1d - 5M post-Dose 2. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, five months (M) post-dose 2 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE (see above) = 6.3, 95% CI 2-sided [-18.0 to 25.7]
Statistical Analysis 3: Comparison: 10PP-HD 2+1d Group vs Synflorix 2+1d Group; VE-10PP-HD 2+1d vs Synflorix 2+1d - 3M post-Dose 3. The analysis aimed to compare occurrences in terms of percentage of subjects with positive nasopharyngeal sample out of the number of subjects with swabs cultured, between 2 groups, three months (M) post-dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; VE (see above) = -3.5, 95% CI 2-sided [-29.3 to 17.2]

7. Secondary Outcome: Number of Subjects With Haematological or Biochemical Abnormalities With Respect to Normal Laboratory Ranges - For Cohort 1/Step 1 Subjects
Description: Assessed biochemical and haematological parameters were: Haemoglobin (Hgb), White cell count (WBC), Platelet counts, Alanine aminotransferase (ALT) and Creatinine (CREA). Per parameter, it was assessed whether subjects had laboratory values below normal, normal, or above normal range. Below = value below the laboratory reference range defined for the specified time point and laboratory parameter. Within = value within the laboratory reference range defined for the specified time point and laboratory parameter. Above = value above the laboratory reference range defined for the specified time point and laboratory parameter. Unknown = value unknown for the specified time point and laboratory parameter. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group
Number analyzed (Participants) | 60 | 60
Participants
  ALT - Status: Unknown | 0 | 0
  ALT - Status: Below | 0 | 0
  ALT - Status: Within | 60 | 57
  ALT - Status: Above | 0 | 3
  CREA - Status: Unknown | 0 | 0
  CREA - Status: Below | 0 | 0
  CREA - Status: Within | 60 | 60
  CREA - Status: Above | 0 | 0
  Hgb - Status: Unknown | 0 | 0
  Hgb - Status: Below | 2 | 2
  Hgb - Status: Within | 57 | 56
  Hgb - Status: Above | 1 | 2
  Platelets - Status: Unknown | 0 | 0
  Platelets - Status: Below | 0 | 0
  Platelets - Status: Within | 59 | 60
  Platelets - Status: Above | 1 | 0
  WBC - Status: Unknown | 0 | 0
  WBC - Status: Below | 0 | 0
  WBC - Status: Within | 60 | 60
  WBC - Status: Above | 0 | 0

8. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - For Step 1/Cohort 1 Subjects
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity. These should also be considered serious: invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation. Any = Occurrence of an SAE, regardless of relationship to vaccination. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: From Day 0 to Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group
Number analyzed (Participants) | 60 | 60
Participants | 0 | 0

9. Secondary Outcome: Antibody Concentrations Against Pneumococcal Pneumolysin Toxoid (Ply) and Pneumococcal Histidine Triad Protein D (PhtD) Proteins - For Cohort 1/Step 1 Subjects
Description: Anti-Ply and anti-PhtD antibody concentrations were measured by Multiplex immunoassay and expressed as geometric mean concentrations (GMCs), in Luminex Units per milliliter (LU/mL). Cut-off of the assay were concentrations higher than or equal to (≥) 599 LU/mL for anti-Ply antibodies and ≥ 391 LU/mL for anti-PhtD antibodies. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity which included all evaluable subjects for whom immunogenicity data were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: LU/mL
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group
Number analyzed (Participants) | 52 | 51
LU/mL
  Anti-Ply | 22794.9 [17570.1 to 29573.3] | 8510.3 [6668.5 to 10860.8]
  Anti-PhtD | 31326.3 [26293.9 to 37321.8] | 16810.0 [13516.3 to 20906.4]

10. Secondary Outcome: Antibody Concentrations Against Protein D (PD) - For Cohort 1/Step 1 Subjects
Description: Anti-PD antibody concentrations were measured by Multiplex immunoassay, expressed as geometric mean concentrations (GMCs), in Luminex Units per milliliter (LU/mL). The cut-off of the assay was an anti-PD antibody concentration higher than or equal to (≥) 112 LU/mL. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: LU/mL
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group
Number analyzed (Participants) | 52 | 51
LU/mL | 137.5 [108.4 to 174.4] | 65.1 [58.2 to 72.8]

11. Secondary Outcome: Antibody Concentrations Against Vaccine Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - For Cohort 1/Step 1 Subjects
Description: Antibody concentrations were measured by 22F-inhibition Enzyme-Linked ImmunoSorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group
Number analyzed (Participants) | 52 | 51
µg/mL
  Anti-1 antibodies | 1.71 [1.33 to 2.22] | 3.12 [2.44 to 4.01]
  Anti-4 antibodies | 4.80 [3.75 to 6.14] | 4.17 [3.33 to 5.21]
  Anti-5 antibodies | 1.17 [0.88 to 1.55] | 1.47 [1.08 to 1.99]
  Anti-6B antibodies | 0.50 [0.34 to 0.73] | 1.57 [0.98 to 2.51]
  Anti-7F antibodies | 2.44 [1.99 to 2.98] | 6.11 [4.44 to 8.41]
  Anti-9V antibodies | 0.89 [0.71 to 1.12] | 2.41 [1.87 to 3.26]
  Anti-14 antibodies | 1.88 [1.39 to 2.53] | 3.77 [2.61 to 5.43]
  Anti-18C antibodies | 7.58 [5.43 to 10.57] | 4.82 [3.46 to 6.71]
  Anti-19F antibodies | 7.82 [5.84 to 10.46] | 5.95 [4.48 to 7.90]
  Anti-23F antibodies | 0.31 [0.21 to 0.46] | 1.11 [0.74 to 1.67]

12. Secondary Outcome: Antibody Concentrations Against Vaccine Serotypes 3, 6A and 19A - For Cohort 1/Step 1 Subjects
Description: as for outcome 11
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group
Number analyzed (Participants) | 52 | 51
µg/mL
  Anti-3 antibodies | 0.25 [0.14 to 0.46] | 2.35 [1.77 to 3.12]
  Anti-6A antibodies | 0.18 [0.12 to 0.27] | 1.36 [0.96 to 1.93]
  Anti-19A antibodies | 1.38 [0.91 to 2.10] | 5.51 [4.02 to 7.55]

13. Secondary Outcome: Antibody Concentrations Against Vaccine Serotype 6C - For Cohort 1/Step 1 Subjects
Description: No analysis was performed on Enzyme-Linked ImmunoSorbent Assay (ELISA) testing for antibody concentrations against vaccine serotype 6C as no specific qualified/validated assay were available. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Arm/Group | 10PP-HD 1D Group | Prevnar13 1D Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - For Cohort 1/Step 1 Subjects
Description: The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 10PP-HD 1d: Group This group consisted in children aged 2-4 years at vaccination enrolled as part of the Cohort 1/Step 1 of the study who received a single dose of the GSK 2189242A (or 10PP) vaccine in its high-dose (HD) formulation at Day 0. The 10PP vaccine was administered intramuscularly in the non-dominant deltoid.
Arm/Group | 10PP-HD 1d | Prevnar 13 1d Group
Number analyzed (Participants) | 52 | 51
Titers
  OPSONO-1: number analyzed (Participants) | 52 | 50
  OPSONO-1 | 17.2 [11.2 to 26.4] | 112.8 [71.9 to 177.0]
  OPSONO-4 | 2818.9 [2009.7 to 3953.8] | 4162.3 [3123.9 to 5545.9]
  OPSONO-5: number analyzed (Participants) | 52 | 49
  OPSONO-5 | 9.0 [6.4 to 12.7] | 89.8 [55.8 to 144.5]
  OPSONO-6B: number analyzed (Participants) | 50 | 51
  OPSONO-6B | 345.3 [171.4 to 695.5] | 5082.5 [3700.2 to 6981.2]
  OPSONO-7F | 6214.0 [5217.1 to 7401.4] | 17781.0 [14034.2 to 22528.0]
  OPSONO-9V | 2880.8 [2264.8 to 3664.5] | 12687.8 [9188.2 to 17520.2]
  OPSONO-14: number analyzed (Participants) | 51 | 51
  OPSONO-14 | 1116.1 [715.5 to 1741.0] | 5985.9 [4313.1 to 8307.4]
  OPSONO-18C: number analyzed (Participants) | 52 | 49
  OPSONO-18C | 3955.4 [3027.7 to 5167.2] | 2799.8 [1931.1 to 4059.2]
  OPSONO-19F | 862.9 [529.2 to 1407.0] | 452.8 [276.2 to 742.2]
  OPSONO-23F: number analyzed (Participants) | 51 | 51
  OPSONO-23F | 2756.7 [1638.0 to 4639.5] | 12652.4 [8076.0 to 19822.2]

15. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotypes 3, 6A and 19A - For Cohort 1/Step 1 Subjects
Description: as for outcome 14
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-HD 1d | Prevnar 13 1d Group
Number analyzed (Participants) | 51 | 51
Titers
  OPSONO-3 | 10.1 [6.5 to 15.8] | 152.5 [120.4 to 193.2]
  OPSONO-6A: number analyzed (Participants) | 47 | 51
  OPSONO-6A | 212.7 [110.4 to 410.0] | 8488.8 [5984.2 to 12041.8]
  OPSONO-19A: number analyzed (Participants) | 49 | 50
  OPSONO-19A | 461.7 [277.2 to 769.0] | 970.3 [701.0 to 1342.9]

16. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotype 6C - For Cohort 1/Step 1 Subjects
Description: No analysis was performed on opsonophagocytic activity for antibody titers against vaccine serotype 6C as no specific qualified/validated assay were available. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Arm/Group | 10PP-HD 1D Group | Prevnar13 1D Group
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Concentrations of Antibodies Inhibiting Pneumococcal Pneumolysin Toxoid (Ply) Haemolysis Activity, or Hem-Ply Antibodies - For Cohort 1/Step 1 Subjects
Description: Concentrations of Hem-Ply antibodies were expressed as geometric mean titers . The cut-off of the assay was an Hem-Ply antibody titer ≥ 140. This outcome concerns subjects enrolled in Cohort 1/Step 1.
Time Frame: At Month 1, or 1 month post vaccination with pneumococcal vaccine (10PP vaccine or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-HD 1d | Prevnar 13 1d Group
Number analyzed (Participants) | 52 | 51
Titers | 682.3 [562.8 to 827.3] | 534.0 [439.4 to 648.9]

18. Secondary Outcome: Antibody Concentrations Against Pneumococcal Pneumolysin Toxoid (Ply) and Pneumococcal Histidine Triad Protein D (PhtD) Proteins - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: Anti-Ply and anti-PhtD antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA) immunoassay and expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). Cut-off of the assay were concentrations higher than or equal to (≥) 12 EL.U/mL for anti-Ply antibodies and ≥ 17 EL.U/mL for anti-PhtD antibodies. This outcome concerns subjects enrolled in Cohort 2/Step 2 who received the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 192 | 195 | 196 | 195
EL.U/mL
  Anti-Ply 1 Mth post dose 3 | 13968.86 [12612.27 to 15471.36] | 16771.16 [15267.84 to 18422.51] | 451.32 [398.68 to 510.91] | 419.47 [377.26 to 466.40]
  Anti-Ply 5 Mth post dose 3: number analyzed (Participants) | 191 | 192 | 195 | 190
  Anti-Ply 5 Mth post dose 3 | 11268.35 [9870.36 to 12864.36] | 10817.78 [9528.87 to 12281.04] | 744.86 [631.27 to 878.89] | 637.49 [539.55 to 753.22]
  Anti-Ply 8 Mth post dose 3: number analyzed (Participants) | 189 | 190 | 195 | 188
  Anti-Ply 8 Mth post dose 3 | 10512.39 [9249.03 to 11948.33] | 10299.57 [9137.48 to 11609.44] | 999.39 [861.41 to 1159.49] | 884.83 [748.83 to 1045.54]
  Anti-PhtD 1 Mth post dose 3 | 2584.28 [2292.67 to 2912.98] | 2188.28 [1934.94 to 2474.80] | 334.18 [292.90 to 381.28] | 486.01 [419.64 to 562.87]
  Anti-PhtD 5 Mth post dose 3: number analyzed (Participants) | 191 | 192 | 195 | 190
  Anti-PhtD 5 Mth post dose 3 | 2242.06 [1971.08 to 2550.29] | 1498.86 [1311.05 to 1713.57] | 936.83 [780.23 to 1124.86] | 1419.77 [1196.01 to 1685.40]
  Anti-PhtD 8 Mth post dose 3: number analyzed (Participants) | 189 | 190 | 195 | 188
  Anti-PhtD 8 Mth post dose 3 | 2608.78 [2318.09 to 2935.92] | 2078.35 [1861.91 to 2319.95] | 1667.91 [1432.09 to 1942.55] | 2380.09 [2118.18 to 2674.39]

19. Secondary Outcome: Antibody Concentrations Against Pneumococcal Pneumolysin Toxoid (Ply) and Pneumococcal Histidine Triad Protein D (PhtD) Proteins - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: Anti-Ply and anti-PhtD antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA) immunoassay and expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). Cut-off of the assay were concentrations higher than or equal to (≥) 12 EL.U/mL for anti-Ply antibodies and ≥ 17 EL.U/mL for anti-PhtD antibodies. This outcome concerns subjects enrolled in Cohort 2/Step 2 who received the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 193 | 193
EL.U/mL
  Anti-Ply 1 Mth post dose 2 | 11491.54 [10168.10 to 12987.23] | 488.79 [427.38 to 559.01]
  Anti-Ply 5 Mth post dose 2: number analyzed (Participants) | 189 | 191
  Anti-Ply 5 Mth post dose 2 | 7453.65 [6460.70 to 8599.21] | 807.67 [676.20 to 964.70]
  Anti-Ply 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-Ply 3 Mth post dose 3 | 17933.07 [15867.00 to 20268.17] | 1114.25 [945.08 to 1313.71]
  Anti-PhtD 1 Mth post dose 2 | 1264.57 [1103.87 to 1448.66] | 368.62 [319.88 to 424.79]
  Anti-PhtD 5 Mth post dose 2: number analyzed (Participants) | 189 | 191
  Anti-PhtD 5 Mth post dose 2 | 1448.08 [1253.08 to 1673.41] | 1036.53 [853.80 to 1258.36]
  Anti-PhtD 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-PhtD 3 Mth post dose 3 | 3250.91 [2956.18 to 3575.02] | 1654.79 [1415.54 to 1934.47]

20. Secondary Outcome: Antibody Concentrations Against Protein D (PD) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: Anti-PD antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA) immunoassay, expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). The cut-off of the assay was anti-PD antibody concentration higher than or equal to (≥) 100 EL.U/mL. This outcome concerns subjects enrolled in Cohort 2/Step 2 who received the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 191 | 193 | 194 | 189
EL.U/mL
  Anti-PD 1 Mth post dose 3: number analyzed (Participants) | 186 | 193 | 187 | 189
  Anti-PD 1 Mth post dose 3 | 1922.8 [1739.3 to 2125.6] | 1833.8 [1628.5 to 2065.0] | 1990.2 [1765.7 to 2243.3] | 84.8 [76.4 to 94.1]
  Anti-PD 5 Mth post dose 3: number analyzed (Participants) | 191 | 191 | 193 | 185
  Anti-PD 5 Mth post dose 3 | 559.2 [496.8 to 629.6] | 499.2 [439.9 to 566.5] | 609.9 [537.0 to 692.8] | 83.1 [74.9 to 92.2]
  Anti-PD 8 Mth post dose 3: number analyzed (Participants) | 187 | 190 | 194 | 187
  Anti-PD 8 Mth post dose 3 | 324.3 [282.2 to 372.7] | 288.2 [248.5 to 334.2] | 344.2 [300.6 to 394.2] | 69.2 [63.6 to 75.3]

21. Secondary Outcome: Antibody Concentrations Against Protein D (PD) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: Anti-PD antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA) immunoassay, expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). The cut-off of the assay was anti-PD antibody concentration higher than or equal to (≥) 100 EL.U/mL. This outcome concerns subjects enrolled in Cohort 2/Step 2 who received the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 190 | 190
EL.U/mL
  Anti-PD 1 Mth post dose 2: number analyzed (Participants) | 187 | 187
  Anti-PD 1 Mth post dose 2 | 990.9 [869.3 to 1129.5] | 1126.7 [999.4 to 1270.2]
  Anti-PD 5 Mth post dose 2: number analyzed (Participants) | 188 | 187
  Anti-PD 5 Mth post dose 2 | 281.3 [247.5 to 319.7] | 313.0 [276.2 to 354.7]
  Anti-PD 3 Mth post dose 3 | 534.8 [468.9 to 610.0] | 664.9 [580.1 to 762.2]

22. Secondary Outcome: Antibody Concentrations Against Vaccine Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - For Cohort 2/Step 2 Subjects Who Received the 3+0 Schedule
Description: Antibody concentrations were measured by 22F-inhibition Enzyme-Linked ImmunoSorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL. This outcome concerns subjects enrolled in Cohort 2/Step 2 who received the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 191 | 195 | 196 | 195
µg/mL
  Anti-1 1 Mth post dose 3: number analyzed (Participants) | 191 | 194 | 193 | 193
  Anti-1 1 Mth post dose 3 | 3.58 [3.17 to 4.03] | 3.20 [2.82 to 3.63] | 3.38 [2.98 to 3.83] | 5.51 [4.92 to 6.17]
  Anti-1 5 Mth post dose 3: number analyzed (Participants) | 190 | 192 | 195 | 189
  Anti-1 5 Mth post dose 3 | 0.67 [0.59 to 0.76] | 0.55 [0.49 to 0.63] | 0.62 [0.55 to 0.71] | 1.16 [1.05 to 1.29]
  Anti-1 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 187
  Anti-1 8 Mth post dose 3 | 0.40 [0.35 to 0.45] | 0.35 [0.31 to 0.40] | 0.40 [0.35 to 0.46] | 0.83 [0.73 to 0.93]
  Anti-4 1 Mth post dose 3: number analyzed (Participants) | 191 | 195 | 195 | 192
  Anti-4 1 Mth post dose 3 | 3.89 [3.43 to 4.41] | 3.15 [2.75 to 3.60] | 3.75 [3.29 to 4.28] | 6.25 [5.63 to 6.93]
  Anti-4 5 Mth post dose 3: number analyzed (Participants) | 191 | 192 | 194 | 190
  Anti-4 5 Mth post dose 3 | 1.19 [1.06 to 1.34] | 1.04 [0.93 to 1.16] | 1.14 [1.00 to 1.29] | 1.06 [0.94 to 1.19]
  Anti-4 8 Mth post dose 3: number analyzed (Participants) | 189 | 190 | 195 | 188
  Anti-4 8 Mth post dose 3 | 0.70 [0.62 to 0.79] | 0.59 [0.52 to 0.68] | 0.66 [0.58 to 0.76] | 0.54 [0.48 to 0.61]
  Anti-5 1 Mth post dose 3: number analyzed (Participants) | 186 | 193 | 187 | 190
  Anti-5 1 Mth post dose 3 | 5.17 [4.54 to 5.88] | 4.83 [4.21 to 5.54] | 5.30 [4.66 to 6.02] | 7.02 [6.14 to 8.02]
  Anti-5 5 Mth post dose 3: number analyzed (Participants) | 190 | 192 | 194 | 190
  Anti-5 5 Mth post dose 3 | 1.37 [1.21 to 1.55] | 1.25 [1.10 to 1.43] | 1.33 [1.17 to 1.51] | 1.79 [1.59 to 2.02]
  Anti-5 8 Mth post dose 3: number analyzed (Participants) | 189 | 187 | 194 | 187
  Anti-5 8 Mth post dose 3 | 0.73 [0.65 to 0.83] | 0.68 [0.59 to 0.79] | 0.69 [0.60 to 0.79] | 1.12 [0.99 to 1.27]
  Anti-6B 1 Mth post dose 3: number analyzed (Participants) | 190 | 194 | 192 | 191
  Anti-6B 1 Mth post dose 3 | 0.91 [0.74 to 1.12] | 0.69 [0.56 to 0.86] | 1.00 [0.80 to 1.25] | 1.35 [1.11 to 1.65]
  Anti-6B 5 Mth post dose 3: number analyzed (Participants) | 190 | 190 | 194 | 189
  Anti-6B 5 Mth post dose 3 | 1.10 [0.94 to 1.29] | 0.86 [0.73 to 1.01] | 1.24 [1.06 to 1.44] | 0.38 [0.33 to 0.44]
  Anti-6B 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 195 | 188
  Anti-6B 8 Mth post dose 3 | 0.87 [0.75 to 1.00] | 0.73 [0.62 to 0.86] | 0.96 [0.83 to 1.11] | 0.29 [0.26 to 0.34]
  Anti-7F 1 Mth post dose 3: number analyzed (Participants) | 190 | 194 | 195 | 195
  Anti-7F 1 Mth post dose 3 | 4.63 [4.10 to 5.22] | 4.10 [3.62 to 4.63] | 4.29 [3.77 to 4.88] | 5.53 [4.96 to 6.17]
  Anti-7F 5 Mth post dose 3: number analyzed (Participants) | 191 | 192 | 195 | 190
  Anti-7F 5 Mth post dose 3 | 2.24 [2.01 to 2.50] | 1.84 [1.63 to 2.08] | 2.19 [1.95 to 2.47] | 2.21 [1.99 to 2.45]
  Anti-7F 8 Mth post dose 3: number analyzed (Participants) | 189 | 190 | 195 | 188
  Anti-7F 8 Mth post dose 3 | 1.54 [1.38 to 1.72] | 1.31 [1.15 to 1.50] | 1.57 [1.39 to 1.78] | 1.65 [1.49 to 1.82]
  Anti-9V 1 Mth post dose 3: number analyzed (Participants) | 188 | 194 | 196 | 194
  Anti-9V 1 Mth post dose 3 | 3.23 [2.83 to 3.68] | 3.25 [2.83 to 3.72] | 3.26 [2.82 to 3.78] | 4.02 [3.45 to 4.69]
  Anti-9V 5 Mth post dose 3: number analyzed (Participants) | 191 | 192 | 193 | 189
  Anti-9V 5 Mth post dose 3 | 1.35 [1.20 to 1.53] | 1.15 [1.02 to 1.30] | 1.33 [1.17 to 1.52] | 0.83 [0.72 to 0.95]
  Anti-9V 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 195 | 188
  Anti-9V 8 Mth post dose 3 | 1.09 [0.95 to 1.25] | 0.87 [0.77 to 1.00] | 1.08 [0.95 to 1.23] | 0.63 [0.55 to 0.73]
  Anti-14 1 Mth post dose 3: number analyzed (Participants) | 191 | 193 | 192 | 194
  Anti-14 1 Mth post dose 3 | 4.36 [3.70 to 5.13] | 4.11 [3.49 to 4.85] | 4.15 [3.52 to 4.89] | 4.66 [3.93 to 5.52]
  Anti-14 5 Mth post dose 3: number analyzed (Participants) | 190 | 192 | 194 | 189
  Anti-14 5 Mth post dose 3 | 2.15 [1.84 to 2.50] | 1.86 [1.56 to 2.22] | 2.13 [1.77 to 2.56] | 3.43 [2.89 to 4.06]
  Anti-14 8 Mth post dose 3: number analyzed (Participants) | 189 | 190 | 195 | 188
  Anti-14 8 Mth post dose 3 | 1.38 [1.18 to 1.61] | 1.37 [1.15 to 1.63] | 1.42 [1.18 to 1.71] | 2.47 [2.10 to 2.92]
  Anti-18C 1 Mth post dose 3: number analyzed (Participants) | 186 | 194 | 189 | 193
  Anti-18C 1 Mth post dose 3 | 15.88 [13.80 to 18.26] | 14.84 [12.88 to 17.09] | 15.66 [13.52 to 18.14] | 5.78 [5.03 to 6.64]
  Anti-18C 5 Mth post dose 3: number analyzed (Participants) | 191 | 192 | 195 | 190
  Anti-18C 5 Mth post dose 3 | 4.09 [3.54 to 4.71] | 3.52 [3.06 to 4.05] | 4.17 [3.60 to 4.83] | 0.95 [0.84 to 1.06]
  Anti-18C 8 Mth post dose 3: number analyzed (Participants) | 189 | 190 | 195 | 188
  Anti-18C 8 Mth post dose 3 | 2.18 [1.90 to 2.51] | 1.82 [1.58 to 2.10] | 2.24 [1.95 to 2.58] | 0.66 [0.58 to 0.75]
  Anti-19F 1 Mth post dose 3: number analyzed (Participants) | 189 | 193 | 193 | 193
  Anti-19F 1 Mth post dose 3 | 9.47 [8.08 to 11.09] | 9.36 [8.04 to 10.91] | 10.04 [8.54 to 11.80] | 5.99 [5.40 to 6.64]
  Anti-19F 5 Mth post dose 3: number analyzed (Participants) | 190 | 191 | 195 | 188
  Anti-19F 5 Mth post dose 3 | 2.65 [2.29 to 3.07] | 2.34 [2.03 to 2.71] | 3.11 [2.67 to 3.62] | 0.96 [0.83 to 1.11]
  Anti-19F 8 Mth post dose 3: number analyzed (Participants) | 189 | 188 | 194 | 187
  Anti-19F 8 Mth post dose 3 | 1.65 [1.40 to 1.93] | 1.45 [1.22 to 1.72] | 1.99 [1.68 to 2.35] | 0.55 [0.46 to 0.66]
  Anti-23F 1 Mth post dose 3: number analyzed (Participants) | 185 | 194 | 189 | 192
  Anti-23F 1 Mth post dose 3 | 1.18 [0.98 to 1.42] | 1.14 [0.95 to 1.38] | 1.22 [0.99 to 1.51] | 2.92 [2.47 to 3.44]
  Anti-23F 5 Mth post dose 3: number analyzed (Participants) | 191 | 192 | 195 | 190
  Anti-23F 5 Mth post dose 3 | 0.78 [0.66 to 0.93] | 0.77 [0.66 to 0.89] | 0.90 [0.77 to 1.06] | 0.47 [0.40 to 0.57]
  Anti-23F 8 Mth post dose 3: number analyzed (Participants) | 189 | 190 | 195 | 188
  Anti-23F 8 Mth post dose 3 | 0.62 [0.53 to 0.73] | 0.59 [0.49 to 0.70] | 0.68 [0.58 to 0.79] | 0.39 [0.31 to 0.48]

23. Secondary Outcome: Antibody Concentrations Against Vaccine Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - For Cohort 2/Step 2 Subjects Who Received the 2+1 Schedule
Description: Antibody concentrations were measured by 22F-inhibition Enzyme-Linked ImmunoSorbent Assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL. This outcome concerns subjects enrolled in Cohort 2/Step 2 who received the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 193 | 193
µg/mL
  Anti-1 1 Mth post dose 2: number analyzed (Participants) | 192 | 191
  Anti-1 1 Mth post dose 2 | 2.52 [2.22 to 2.86] | 2.41 [2.13 to 2.72]
  Anti-1 5 Mth post dose 2: number analyzed (Participants) | 189 | 191
  Anti-1 5 Mth post dose 2 | 0.44 [0.39 to 0.49] | 0.42 [0.37 to 0.48]
  Anti-1 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-1 3 Mth post dose 3 | 1.65 [1.43 to 1.90] | 1.61 [1.41 to 1.83]
  Anti-4 1 Mth post dose 2: number analyzed (Participants) | 192 | 193
  Anti-4 1 Mth post dose 2 | 2.79 [2.42 to 3.22] | 2.67 [2.30 to 3.09]
  Anti-4 5 Mth post dose 2: number analyzed (Participants) | 189 | 190
  Anti-4 5 Mth post dose 2 | 0.79 [0.70 to 0.89] | 0.76 [0.67 to 0.86]
  Anti-4 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-4 3 Mth post dose 3 | 2.15 [1.91 to 2.42] | 1.92 [1.71 to 2.16]
  Anti-5 1 Mth post dose 2: number analyzed (Participants) | 188 | 186
  Anti-5 1 Mth post dose 2 | 3.74 [3.29 to 4.26] | 3.40 [2.96 to 3.91]
  Anti-5 5 Mth post dose 2: number analyzed (Participants) | 188 | 190
  Anti-5 5 Mth post dose 2 | 1.07 [0.95 to 1.21] | 0.92 [0.81 to 1.04]
  Anti-5 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-5 3 Mth post dose 3 | 2.86 [2.53 to 3.23] | 2.34 [2.04 to 2.69]
  Anti-6B 1 Mth post dose 2: number analyzed (Participants) | 189 | 189
  Anti-6B 1 Mth post dose 2 | 0.51 [0.40 to 0.64] | 0.51 [0.41 to 0.64]
  Anti-6B 5 Mth post dose 2: number analyzed (Participants) | 186 | 189
  Anti-6B 5 Mth post dose 2 | 0.63 [0.53 to 0.75] | 0.67 [0.58 to 0.79]
  Anti-6B 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-6B 3 Mth post dose 3 | 1.35 [1.17 to 1.56] | 1.39 [1.21 to 1.61]
  Anti-7F 1 Mth post dose 2: number analyzed (Participants) | 192 | 191
  Anti-7F 1 Mth post dose 2 | 3.29 [2.95 to 3.67] | 3.06 [2.68 to 3.49]
  Anti-7F 5 Mth post dose 2: number analyzed (Participants) | 189 | 191
  Anti-7F 5 Mth post dose 2 | 1.47 [1.30 to 1.66] | 1.48 [1.30 to 1.68]
  Anti-7F 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-7F 3 Mth post dose 3 | 3.36 [3.00 to 3.77] | 3.40 [3.04 to 3.81]
  Anti-9V 1 Mth post dose 2: number analyzed (Participants) | 191 | 191
  Anti-9V 1 Mth post dose 2 | 1.85 [1.60 to 2.14] | 1.97 [1.72 to 2.26]
  Anti-9V 5 Mth post dose 2: number analyzed (Participants) | 189 | 191
  Anti-9V 5 Mth post dose 2 | 0.85 [0.75 to 0.95] | 0.81 [0.72 to 0.91]
  Anti-9V 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-9V 3 Mth post dose 3 | 2.86 [2.54 to 3.23] | 2.67 [2.32 to 3.06]
  Anti-14 1 Mth post dose 2: number analyzed (Participants) | 192 | 190
  Anti-14 1 Mth post dose 2 | 2.39 [2.01 to 2.85] | 2.29 [1.92 to 2.72]
  Anti-14 5 Mth post dose 2: number analyzed (Participants) | 189 | 191
  Anti-14 5 Mth post dose 2 | 0.85 [0.70 to 1.03] | 0.89 [0.75 to 1.06]
  Anti-14 3 Mth post dose 3: number analyzed (Participants) | 190 | 189
  Anti-14 3 Mth post dose 3 | 2.40 [2.07 to 2.79] | 2.42 [2.09 to 2.80]
  Anti-18C 1 Mth post dose 2: number analyzed (Participants) | 191 | 188
  Anti-18C 1 Mth post dose 2 | 11.33 [9.39 to 13.68] | 10.88 [8.98 to 13.18]
  Anti-18C 5 Mth post dose 2: number analyzed (Participants) | 189 | 190
  Anti-18C 5 Mth post dose 2 | 3.00 [2.54 to 3.53] | 3.18 [2.71 to 3.74]
  Anti-18C 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-18C 3 Mth post dose 3 | 18.38 [15.94 to 21.19] | 16.24 [14.11 to 18.69]
  Anti-19F 1 Mth post dose 2: number analyzed (Participants) | 193 | 192
  Anti-19F 1 Mth post dose 2 | 7.33 [6.17 to 8.71] | 7.85 [6.61 to 9.32]
  Anti-19F 5 Mth post dose 2: number analyzed (Participants) | 187 | 191
  Anti-19F 5 Mth post dose 2 | 2.38 [2.07 to 2.74] | 2.48 [2.12 to 2.90]
  Anti-19F 3 Mth post dose 3: number analyzed (Participants) | 189 | 189
  Anti-19F 3 Mth post dose 3 | 5.99 [5.13 to 7.01] | 6.27 [5.36 to 7.32]
  Anti-23F 1 Mth post dose 2: number analyzed (Participants) | 189 | 189
  Anti-23F 1 Mth post dose 2 | 0.63 [0.51 to 0.78] | 0.67 [0.53 to 0.84]
  Anti-23F 5 Mth post dose 2: number analyzed (Participants) | 189 | 191
  Anti-23F 5 Mth post dose 2 | 0.44 [0.37 to 0.52] | 0.46 [0.39 to 0.55]
  Anti-23F 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-23F 3 Mth post dose 3 | 1.46 [1.24 to 1.72] | 1.50 [1.27 to 1.76]

24. Secondary Outcome: Antibody Concentrations Against Vaccine Serotypes 3 and 19A - For Cohort 2/Step 2 Subjects Who Received the 3+0 Schedule
Description: as for outcome 22
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 189 | 192 | 195 | 192
µg/mL
  Anti-3 1 Mth post dose 3: number analyzed (Participants) | 184 | 192 | 186 | 192
  Anti-3 1 Mth post dose 3 | 0.05 [0.04 to 0.06] | 0.05 [0.04 to 0.05] | 0.05 [0.04 to 0.06] | 4.52 [4.15 to 4.92]
  Anti-3 5 Mth post dose 3: number analyzed (Participants) | 189 | 192 | 191 | 188
  Anti-3 5 Mth post dose 3 | 0.06 [0.05 to 0.07] | 0.06 [0.05 to 0.08] | 0.07 [0.06 to 0.09] | 0.60 [0.52 to 0.68]
  Anti-3 8 Mth post dose 3: number analyzed (Participants) | 188 | 190 | 195 | 187
  Anti-3 8 Mth post dose 3 | 0.08 [0.07 to 0.11] | 0.09 [0.07 to 0.12] | 0.09 [0.07 to 0.11] | 0.32 [0.27 to 0.38]
  Anti-19A 1 Mth post dose 3: number analyzed (Participants) | 185 | 190 | 182 | 191
  Anti-19A 1 Mth post dose 3 | 0.24 [0.20 to 0.29] | 0.20 [0.17 to 0.24] | 0.23 [0.19 to 0.27] | 5.27 [4.41 to 6.30]
  Anti-19A 5 Mth post dose 3: number analyzed (Participants) | 187 | 186 | 194 | 187
  Anti-19A 5 Mth post dose 3 | 0.21 [0.17 to 0.25] | 0.17 [0.14 to 0.21] | 0.24 [0.20 to 0.30] | 0.91 [0.76 to 1.08]
  Anti-19A 8 Mth post dose 3: number analyzed (Participants) | 184 | 185 | 192 | 185
  Anti-19A 8 Mth post dose 3 | 0.24 [0.19 to 0.29] | 0.21 [0.17 to 0.27] | 0.27 [0.22 to 0.34] | 0.64 [0.52 to 0.79]

25. Secondary Outcome: Antibody Concentrations Against Vaccine Serotypes 3 and 19A - For Cohort 2/Step 2 Subjects Who Received the 2+1 Schedule
Description: as for outcome 23
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 190 | 191
µg/mL
  Anti-3 1 Mth post dose 2: number analyzed (Participants) | 186 | 187
  Anti-3 1 Mth post dose 2 | 0.04 [0.04 to 0.05] | 0.05 [0.04 to 0.06]
  Anti-3 5 Mth post dose 2: number analyzed (Participants) | 187 | 191
  Anti-3 5 Mth post dose 2 | 0.06 [0.05 to 0.07] | 0.07 [0.05 to 0.09]
  Anti-3 3 Mth post dose 3: number analyzed (Participants) | 190 | 190
  Anti-3 3 Mth post dose 3 | 0.07 [0.06 to 0.09] | 0.08 [0.06 to 0.10]
  Anti-19A 1 Mth post dose 2: number analyzed (Participants) | 187 | 186
  Anti-19A 1 Mth post dose 2 | 0.24 [0.20 to 0.29] | 0.25 [0.20 to 0.30]
  Anti-19A 5 Mth post dose 2: number analyzed (Participants) | 183 | 190
  Anti-19A 5 Mth post dose 2 | 0.18 [0.15 to 0.22] | 0.19 [0.15 to 0.24]
  Anti-19A 3 Mth post dose 3: number analyzed (Participants) | 190 | 187
  Anti-19A 3 Mth post dose 3 | 0.56 [0.43 to 0.71] | 0.64 [0.50 to 0.81]

26. Secondary Outcome: Antibody Concentrations Against Vaccine Serotype 6A - For Cohort 2/Step 2 Subjects Who Received the 3+0 Schedule
Description: as for outcome 22
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 190 | 192 | 192 | 190
µg/mL
  Anti-6A 1Mth post dose 3: number analyzed (Participants) | 185 | 192 | 187 | 190
  Anti-6A 1Mth post dose 3 | 0.13 [0.11 to 0.16] | 0.13 [0.11 to 0.15] | 0.13 [0.11 to 0.15] | 3.01 [2.60 to 3.48]
  Anti-6A 5 Mth post dose 3: number analyzed (Participants) | 190 | 190 | 192 | 189
  Anti-6A 5 Mth post dose 3 | 0.17 [0.14 to 0.20] | 0.15 [0.13 to 0.18] | 0.22 [0.18 to 0.27] | 1.0 [0.89 to 1.13]
  Anti-6A 8 Mth post dose 3: number analyzed (Participants) | 177 | 179 | 178 | 148
  Anti-6A 8 Mth post dose 3 | 0.16 [0.14 to 0.19] | 0.15 [0.13 to 0.18] | 0.18 [0.15 to 0.22] | 0.59 [0.51 to 0.68]

27. Secondary Outcome: Antibody Concentrations Against Vaccine Serotype 6A - For Cohort 2/Step 2 Subjects Who Received the 2+1 Schedule
Description: as for outcome 23
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 187 | 189
µg/mL
  Anti-6A 1 Mth post dose 2: number analyzed (Participants) | 187 | 187
  Anti-6A 1 Mth post dose 2 | 0.11 [0.09 to 0.12] | 0.11 [0.09 to 0.13]
  Anti-6A 5 Mth post-dose 2: number analyzed (Participants) | 185 | 189
  Anti-6A 5 Mth post-dose 2 | 0.10 [0.09 to 0.12] | 0.12 [0.10 to 0.14]
  Anti-6A 3 Mth post dose 3: number analyzed (Participants) | 174 | 175
  Anti-6A 3 Mth post dose 3 | 0.14 [0.12 to 0.16] | 0.15 [0.12 to 0.17]

28. Secondary Outcome: Antibody Concentrations Against Vaccine Serotype 6C - For Cohort 2/Step 2 Subjects Who Received the 3+0 Schedule
Description: No analysis was performed on Enzyme-Linked ImmunoSorbent Assay (ELISA) testing for antibody concentrations against vaccine serotype 6C as no specific qualified/validated assay was available. This outcome concerns subjects enrolled in Cohort 2/Step 2.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

29. Secondary Outcome: Antibody Concentrations Against Vaccine Serotype 6C - For Cohort 2/Step 2 Subjects Who Received the 2+1 Schedule
Description: as for outcome 28
Time Frame: as for outcome 6
Population: as for outcome 9
Arm/Group | 10PP-HD 2+1D Group | Synflorix 2+1D Group
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 93 | 96 | 98 | 96
Titers
  OPSONO-1 1 Mth post dose 3 | 136.3 [98.8 to 188.0] | 62.7 [42.8 to 91.9] | 109.9 [79.2 to 152.6] | 161.4 [116.5 to 223.8]
  OPSONO-1 5 Mth post dose 3: number analyzed (Participants) | 93 | 95 | 94 | 90
  OPSONO-1 5 Mth post dose 3 | 14.1 [9.9 to 20.0] | 10.1 [7.4 to 13.8] | 11.0 [7.9 to 15.3] | 14.3 [9.9 to 20.4]
  OPSONO-1 8 Mth post dose 3: number analyzed (Participants) | 91 | 95 | 96 | 88
  OPSONO-1 8 Mth post dose 3 | 10.0 [7.3 to 13.6] | 8.4 [6.4 to 11.0] | 9.3 [6.9 to 12.5] | 12.5 [8.8 to 17.6]
  OPSONO-4 1 Mth post dose 3: number analyzed (Participants) | 91 | 95 | 98 | 94
  OPSONO-4 1 Mth post dose 3 | 835.0 [657.1 to 1061.0] | 784.0 [633.1 to 970.8] | 715.6 [586.5 to 873.2] | 1022.7 [839.6 to 1245.7]
  OPSONO-4 5 Mth post dose 3: number analyzed (Participants) | 86 | 91 | 93 | 84
  OPSONO-4 5 Mth post dose 3 | 86.0 [58.5 to 126.4] | 48.2 [31.5 to 73.7] | 54.7 [37.2 to 80.4] | 62.8 [40.0 to 98.4]
  OPSONO-4 8 Mth post dose 3: number analyzed (Participants) | 86 | 90 | 91 | 85
  OPSONO-4 8 Mth post dose 3 | 48.2 [31.0 to 74.9] | 34.3 [21.8 to 53.9] | 41.7 [27.4 to 63.7] | 41.8 [25.9 to 67.5]
  OPSONO-5 1 Mth post dose 3: number analyzed (Participants) | 93 | 95 | 97 | 96
  OPSONO-5 1 Mth post dose 3 | 97.9 [75.5 to 127.0] | 51.4 [37.8 to 70.1] | 76.7 [58.5 to 100.6] | 91.5 [69.7 to 120.2]
  OPSONO-5 5 Mth post dose 3: number analyzed (Participants) | 93 | 96 | 97 | 90
  OPSONO-5 5 Mth post dose 3 | 19.7 [14.9 to 26.1] | 13.1 [10.0 to 17.3] | 16.2 [12.1 to 21.5] | 17.4 [13.2 to 23.0]
  OPSONO-5 8 Mth post dose 3: number analyzed (Participants) | 92 | 95 | 98 | 89
  OPSONO-5 8 Mth post dose 3 | 9.4 [7.4 to 11.9] | 8.3 [6.5 to 10.5] | 11.2 [8.7 to 14.2] | 10.8 [8.5 to 13.6]
  OPSONO-6B 1 Mth post dose 3: number analyzed (Participants) | 93 | 95 | 96 | 96
  OPSONO-6B 1 Mth post dose 3 | 827.6 [601.4 to 1138.9] | 432.8 [293.1 to 638.8] | 814.6 [594.1 to 1116.9] | 1317.6 [937.1 to 1852.6]
  OPSONO-6B 5 Mth post dose 3: number analyzed (Participants) | 93 | 91 | 97 | 88
  OPSONO-6B 5 Mth post dose 3 | 242.4 [158.9 to 369.9] | 251.3 [169.1 to 373.4] | 324.0 [227.2 to 461.9] | 90.9 [53.3 to 155.0]
  OPSONO-6B 8 Mth post dose 3: number analyzed (Participants) | 90 | 88 | 97 | 83
  OPSONO-6B 8 Mth post dose 3 | 146.9 [95.9 to 225.1] | 126.0 [80.4 to 197.4] | 233.1 [160.7 to 338.1] | 73.7 [43.3 to 125.4]
  OPSONO-7F 1 Mth post dose 3: number analyzed (Participants) | 93 | 95 | 98 | 96
  OPSONO-7F 1 Mth post dose 3 | 3755.3 [3060.5 to 4607.9] | 2993.3 [2440.1 to 3672.0] | 3767.9 [2981.2 to 4762.1] | 7241.0 [5923.2 to 8852.1]
  OPSONO-7F 5 Mth post dose 3: number analyzed (Participants) | 93 | 96 | 97 | 90
  OPSONO-7F 5 Mth post dose 3 | 2072.1 [1634.8 to 2626.3] | 1850.6 [1454.8 to 2354.1] | 1710.3 [1329.7 to 2199.9] | 3652.1 [2878.1 to 4634.2]
  OPSONO-7F 8 Mth post dose 3: number analyzed (Participants) | 92 | 95 | 98 | 89
  OPSONO-7F 8 Mth post dose 3 | 2001.5 [1629.3 to 2458.7] | 2313.0 [1851.4 to 2889.8] | 2291.2 [1903.9 to 2757.3] | 3054.1 [2502.7 to 3727.0]
  OPSONO-9V 1 Mth post dose 3: number analyzed (Participants) | 93 | 96 | 98 | 94
  OPSONO-9V 1 Mth post dose 3 | 909.2 [722.3 to 1144.5] | 1113.1 [888.0 to 1395.3] | 1044.6 [788.6 to 1383.6] | 878.3 [647.7 to 1191.0]
  OPSONO-9V 5 Mth post dose 3: number analyzed (Participants) | 92 | 95 | 97 | 90
  OPSONO-9V 5 Mth post dose 3 | 360.3 [253.2 to 512.7] | 449.2 [347.2 to 581.3] | 320.1 [236.2 to 433.6] | 342.8 [240.3 to 489.0]
  OPSONO-9V 8 Mth post dose 3: number analyzed (Participants) | 89 | 92 | 97 | 88
  OPSONO-9V 8 Mth post dose 3 | 330.6 [230.2 to 474.9] | 436.7 [322.5 to 591.4] | 277.0 [196.1 to 391.4] | 308.6 [216.6 to 439.7]
  OPSONO-14 1 Mth post dose 3: number analyzed (Participants) | 93 | 95 | 97 | 93
  OPSONO-14 1 Mth post dose 3 | 1176.2 [823.1 to 1680.9] | 1169.8 [845.3 to 1618.9] | 1139.9 [773.2 to 1680.4] | 2504.7 [1665.7 to 3766.3]
  OPSONO-14 5 Mth post dose 3: number analyzed (Participants) | 89 | 95 | 95 | 89
  OPSONO-14 5 Mth post dose 3 | 188.9 [129.7 to 275.0] | 181.3 [125.6 to 261.5] | 233.4 [160.2 to 340.1] | 499.3 [350.5 to 711.1]
  OPSONO-14 8 Mth post dose 3: number analyzed (Participants) | 88 | 89 | 95 | 89
  OPSONO-14 8 Mth post dose 3 | 152.9 [103.0 to 227.1] | 186.9 [130.5 to 267.6] | 223.1 [159.0 to 313.2] | 371.0 [257.6 to 534.2]
  OPSONO-18C 1 Mth post dose 3: number analyzed (Participants) | 93 | 96 | 98 | 94
  OPSONO-18C 1 Mth post dose 3 | 666.2 [542.9 to 817.6] | 532.0 [413.8 to 683.9] | 623.6 [493.1 to 788.6] | 277.7 [209.9 to 367.5]
  OPSONO-18C 5 Mth post dose 3: number analyzed (Participants) | 92 | 95 | 96 | 90
  OPSONO-18C 5 Mth post dose 3 | 39.8 [29.4 to 54.0] | 32.0 [22.9 to 44.6] | 44.1 [32.7 to 59.5] | 9.1 [7.0 to 11.8]
  OPSONO-18C 8 Mth post dose 3: number analyzed (Participants) | 88 | 92 | 97 | 88
  OPSONO-18C 8 Mth post dose 3 | 13.6 [10.2 to 18.1] | 11.7 [9.0 to 15.1] | 16.9 [12.8 to 22.4] | 6.5 [5.0 to 8.3]
  OPSONO-19F 1 Mth post dose 3: number analyzed (Participants) | 90 | 95 | 98 | 94
  OPSONO-19F 1 Mth post dose 3 | 420.3 [307.6 to 574.2] | 340.6 [242.7 to 478.0] | 518.3 [389.1 to 690.4] | 84.8 [66.1 to 108.9]
  OPSONO-19F 5 Mth post dose 3: number analyzed (Participants) | 92 | 96 | 98 | 91
  OPSONO-19F 5 Mth post dose 3 | 47.2 [35.3 to 62.9] | 30.7 [22.8 to 41.4] | 66.9 [49.3 to 90.9] | 7.2 [5.4 to 9.5]
  OPSONO-19F 8 Mth post dose 3: number analyzed (Participants) | 92 | 94 | 97 | 89
  OPSONO-19F 8 Mth post dose 3 | 22.0 [16.3 to 29.6] | 20.3 [14.6 to 28.5] | 32.5 [23.6 to 44.7] | 7.0 [5.4 to 9.2]
  OPSONO-23F 1 Mth post dose 3: number analyzed (Participants) | 93 | 94 | 98 | 96
  OPSONO-23F 1 Mth post dose 3 | 1421.3 [976.4 to 2068.9] | 965.1 [622.7 to 1495.8] | 1030.2 [693.0 to 1531.4] | 2821.9 [1913.1 to 4162.3]
  OPSONO-23F 5 Mth post dose 3: number analyzed (Participants) | 85 | 87 | 90 | 86
  OPSONO-23F 5 Mth post dose 3 | 307.4 [183.0 to 516.3] | 387.1 [234.4 to 639.1] | 239.5 [140.2 to 409.1] | 638.6 [369.2 to 1104.6]
  OPSONO-23F 8 Mth post dose 3: number analyzed (Participants) | 87 | 81 | 89 | 83
  OPSONO-23F 8 Mth post dose 3 | 306.2 [172.3 to 543.9] | 385.9 [221.1 to 673.5] | 410.8 [246.7 to 684.2] | 650.4 [367.1 to 1152.3]

31. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 10PP-HD 2+1d Group: This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received the GSK 2189242A (or 10PP) vaccine, in its high-dose (HD) formulation, and EPI vaccines according to a 2+1 Schedule. That is, subjects received 2 doses of the 10PP vaccine, HD formulation co-administered with Tritanrix™-Hep B/Hib and Polio Sabin™ at 2-4 months of age (at Day 0 and Month 2), followed by a third dose of the same formulation co-administered with M-Vac™, Stamaril™ and Polio Sabin™ at approximately 9 months of age. The 2nd doses of Tritanrix™-Hep B/Hib and Polio Sabin™ in EPI vaccines were administered without any pneumococcal vaccine at 3 months of age. The 10PP vaccine was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 98 | 97
Titers
  OPSONO-1 1 Mth post dose 2 | 67.3 [46.5 to 97.4] | 58.0 [40.4 to 83.4]
  OPSONO-1 5 Mth post dose 2: number analyzed (Participants) | 95 | 95
  OPSONO-1 5 Mth post dose 2 | 7.7 [6.0 to 9.8] | 8.1 [6.1 to 10.7]
  OPSONO-1 3 Mth post dose 3: number analyzed (Participants) | 95 | 95
  OPSONO-1 3 Mth post dose 3 | 58.8 [38.2 to 90.7] | 57.5 [37.8 to 87.5]
  OPSONO-4 1 Mth post dose 2: number analyzed (Participants) | 97 | 96
  OPSONO-4 1 Mth post dose 2 | 461.9 [377.9 to 564.5] | 427.2 [327.0 to 558.0]
  OPSONO-4 5 Mth post dose 2: number analyzed (Participants) | 92 | 90
  OPSONO-4 5 Mth post dose 2 | 27.0 [18.6 to 39.2] | 27.4 [18.6 to 40.4]
  OPSONO-4 3 Mth post dose 3: number analyzed (Participants) | 93 | 91
  OPSONO-4 3 Mth post dose 3 | 260.0 [190.0 to 355.8] | 241.1 [170.4 to 341.0]
  OPSONO-5 1 Mth post dose 2 | 49.1 [37.0 to 65.0] | 49.1 [36.2 to 66.6]
  OPSONO-5 5 Mth post dose 2: number analyzed (Participants) | 95 | 95
  OPSONO-5 5 Mth post dose 2 | 11.8 [9.3 to 15.1] | 12.6 [9.7 to 16.4]
  OPSONO-5 3 Mth post dose 3: number analyzed (Participants) | 96 | 95
  OPSONO-5 3 Mth post dose 3 | 58.2 [44.0 to 77.0] | 47.0 [34.4 to 64.2]
  OPSONO-6B 1 Mth post dose 2: number analyzed (Participants) | 95 | 96
  OPSONO-6B 1 Mth post dose 2 | 359.8 [240.2 to 539.0] | 331.7 [223.1 to 493.2]
  OPSONO-6B 5 Mth post dose 2: number analyzed (Participants) | 91 | 91
  OPSONO-6B 5 Mth post dose 2 | 159.1 [102.0 to 248.0] | 111.1 [68.3 to 180.7]
  OPSONO-6B 3 Mth post dose 3: number analyzed (Participants) | 94 | 89
  OPSONO-6B 3 Mth post dose 3 | 214.7 [146.2 to 315.1] | 192.0 [130.0 to 283.6]
  OPSONO-7F 1 Mth post dose 2: number analyzed (Participants) | 98 | 96
  OPSONO-7F 1 Mth post dose 2 | 2643.3 [2122.6 to 3291.6] | 2336.3 [1923.9 to 2837.3]
  OPSONO-7F 5 Mth post dose 2: number analyzed (Participants) | 95 | 94
  OPSONO-7F 5 Mth post dose 2 | 1258.2 [972.6 to 1627.6] | 1466.4 [1150.1 to 1869.7]
  OPSONO-7F 3 Mth post dose 3: number analyzed (Participants) | 96 | 95
  OPSONO-7F 3 Mth post dose 3 | 2767.6 [2261.7 to 3386.7] | 2963.6 [2379.0 to 3691.9]
  OPSONO-9V 1 Mth post dose 2: number analyzed (Participants) | 98 | 96
  OPSONO-9V 1 Mth post dose 2 | 783.7 [609.0 to 1008.5] | 763.2 [625.4 to 931.4]
  OPSONO-9V 5 Mth post dose 2: number analyzed (Participants) | 91 | 94
  OPSONO-9V 5 Mth post dose 2 | 241.3 [159.0 to 366.2] | 163.3 [113.8 to 234.3]
  OPSONO-9V 3 Mth post dose 3: number analyzed (Participants) | 95 | 95
  OPSONO-9V 3 Mth post dose 3 | 1044.3 [818.8 to 1332.0] | 712.4 [534.2 to 950.0]
  OPSONO-14 1 Mth post dose 2: number analyzed (Participants) | 98 | 96
  OPSONO-14 1 Mth post dose 2 | 349.7 [231.7 to 527.8] | 310.5 [200.1 to 481.9]
  OPSONO-14 5 Mth post dose 2: number analyzed (Participants) | 89 | 91
  OPSONO-14 5 Mth post dose 2 | 54.3 [35.5 to 83.0] | 40.2 [26.6 to 60.8]
  OPSONO-14 3 Mth post dose 3: number analyzed (Participants) | 93 | 93
  OPSONO-14 3 Mth post dose 3 | 335.9 [257.2 to 438.7] | 254.6 [180.4 to 359.4]
  OPSONO-18C 1 Mth post dose 2 | 464.7 [317.0 to 681.2] | 459.7 [330.7 to 639.1]
  OPSONO-18C 5 Mth post dose 2: number analyzed (Participants) | 93 | 95
  OPSONO-18C 5 Mth post dose 2 | 28.4 [20.3 to 39.7] | 33.6 [23.5 to 47.8]
  OPSONO-18C 3 Mth post dose 3: number analyzed (Participants) | 96 | 94
  OPSONO-18C 3 Mth post dose 3 | 562.8 [405.0 to 782.0] | 522.0 [390.0 to 698.7]
  OPSONO-19F 1 Mth post dose 2: number analyzed (Participants) | 96 | 96
  OPSONO-19F 1 Mth post dose 2 | 299.3 [213.5 to 419.6] | 284.7 [201.1 to 403.1]
  OPSONO-19F 5 Mth post dose 2: number analyzed (Participants) | 93 | 94
  OPSONO-19F 5 Mth post dose 2 | 35.5 [26.0 to 48.3] | 38.7 [27.6 to 54.3]
  OPSONO-19F 3 Mth post dose 3: number analyzed (Participants) | 96 | 95
  OPSONO-19F 3 Mth post dose 3 | 203.6 [140.5 to 295.1] | 168.1 [110.0 to 256.8]
  OPSONO-23F 1 Mth post dose 2: number analyzed (Participants) | 94 | 95
  OPSONO-23F 1 Mth post dose 2 | 539.6 [343.1 to 848.6] | 493.9 [308.8 to 789.8]
  OPSONO-23F 5 Mth post dose 2: number analyzed (Participants) | 90 | 91
  OPSONO-23F 5 Mth post dose 2 | 156.5 [88.7 to 276.3] | 158.6 [91.1 to 276.1]
  OPSONO-23F 3 Mth post dose 3: number analyzed (Participants) | 95 | 91
  OPSONO-23F 3 Mth post dose 3 | 612.2 [395.6 to 947.4] | 835.7 [548.1 to 1274.1]

32. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotypes 3 and 6A - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: as for outcome 30
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 92 | 94 | 97 | 96
Titers
  OPSONO-3 1 Mth post dose 3: number analyzed (Participants) | 92 | 92 | 97 | 96
  OPSONO-3 1 Mth post dose 3 | 5.3 [4.3 to 6.4] | 4.5 [4.0 to 5.1] | 4.8 [4.2 to 5.5] | 98.3 [82.8 to 116.7]
  OPSONO-3 5 Mth post dose 3: number analyzed (Participants) | 91 | 94 | 94 | 89
  OPSONO-3 5 Mth post dose 3 | 7.1 [5.6 to 9.0] | 5.5 [4.5 to 6.6] | 6.7 [5.3 to 8.5] | 15.1 [11.0 to 20.6]
  OPSONO-3 8 Mth post dose 3: number analyzed (Participants) | 86 | 91 | 95 | 87
  OPSONO-3 8 Mth post dose 3 | 8.1 [6.3 to 10.5] | 8.3 [6.3 to 11.0] | 7.8 [6.1 to 10.1] | 12.3 [9.0 to 16.7]
  OPSONO-6A 1 Mth post dose 3: number analyzed (Participants) | 88 | 91 | 96 | 96
  OPSONO-6A 1 Mth post dose 3 | 13.7 [9.0 to 20.9] | 11.8 [8.0 to 17.4] | 11.3 [7.7 to 16.5] | 2770.0 [2216.1 to 3462.4]
  OPSONO-6A 5 Mth post dose 3: number analyzed (Participants) | 92 | 92 | 94 | 88
  OPSONO-6A 5 Mth post dose 3 | 14.8 [9.5 to 23.2] | 12.0 [8.0 to 17.9] | 20.2 [12.7 to 32.0] | 602.0 [433.4 to 836.2]
  OPSONO-6A 8 Mth post dose 3: number analyzed (Participants) | 86 | 86 | 88 | 87
  OPSONO-6A 8 Mth post dose 3 | 14.8 [9.4 to 23.3] | 12.4 [8.1 to 19.1] | 18.5 [11.7 to 29.3] | 260.1 [167.4 to 404.2]

33. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotypes 3 and 6A - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: as for outcome 31
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 96 | 97
Titers
  OPSONO-3 1 Mth post dose 2 | 4.7 [4.2 to 5.4] | 5.1 [4.2 to 6.1]
  OPSONO-3 5 Mth post dose 2: number analyzed (Participants) | 87 | 86
  OPSONO-3 5 Mth post dose 2 | 5.9 [4.8 to 7.3] | 5.9 [4.6 to 7.6]
  OPSONO-3 3 Mth post dose 3: number analyzed (Participants) | 92 | 93
  OPSONO-3 3 Mth post dose 3 | 7.4 [5.7 to 9.6] | 6.8 [5.4 to 8.4]
  OPSONO-6A 1 Mth post dose 2 | 6.7 [5.1 to 8.8] | 6.7 [5.1 to 8.7]
  OPSONO-6A 5 Mth post dose 2: number analyzed (Participants) | 93 | 95
  OPSONO-6A 5 Mth post dose 2 | 12.4 [8.4 to 18.3] | 12.2 [8.2 to 18.3]
  OPSONO-6A 3 Mth post dose 3: number analyzed (Participants) | 88 | 91
  OPSONO-6A 3 Mth post dose 3 | 12.6 [8.3 to 19.2] | 10.0 [6.7 to 15.0]

34. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotype 19A - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) to the serotype-specific Lower Limit of Quantification ( = 143). This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 71 | 79 | 71 | 89
Titers
  OPSONO-19A 1 Mth post dose 3: number analyzed (Participants) | 70 | 72 | 71 | 89
  OPSONO-19A 1 Mth post dose 3 | 347.0 [238.0 to 505.9] | 281.1 [192.8 to 409.8] | 369.8 [257.5 to 531.0] | 2652.8 [2277.5 to 3089.9]
  OPSONO-19A 5 Mth post dose 3: number analyzed (Participants) | 71 | 75 | 61 | 69
  OPSONO-19A 5 Mth post dose 3 | 120.4 [91.9 to 157.8] | 121.6 [94.3 to 156.8] | 140.2 [102.1 to 192.4] | 704.2 [498.5 to 994.8]
  OPSONO-19A 8 Mth post dose 3: number analyzed (Participants) | 67 | 79 | 69 | 60
  OPSONO-19A 8 Mth post dose 3 | 155.2 [109.1 to 220.9] | 151.5 [110.0 to 208.7] | 138.7 [101.3 to 190.0] | 394.4 [261.8 to 594.2]

35. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotype 19A - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) to the serotype-specific Lower Limit of Quantification ( = 143). This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 72 | 81
Titers
  OPSONO-19A 1 Mth post dose 2: number analyzed (Participants) | 69 | 71
  OPSONO-19A 1 Mth post dose 2 | 231.3 [164.5 to 325.4] | 177.4 [129.4 to 243.2]
  OPSONO-19A 5 Mth post dose 2: number analyzed (Participants) | 67 | 81
  OPSONO-19A 5 Mth post dose 2 | 99.1 [80.0 to 122.7] | 107.4 [84.5 to 136.5]
  OPSONO-19A 3 Mth post dose 3: number analyzed (Participants) | 72 | 79
  OPSONO-19A 3 Mth post dose 3 | 274.2 [187.6 to 400.8] | 361.2 [247.5 to 527.2]

36. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotype 6C - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: No analysis was performed on opsonophagocytic activity for antibody titers against vaccine serotype 6C as no specific qualified/validated assay was available. This outcome concerns subjects enrolled in Cohort 2/Step 2.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

37. Secondary Outcome: Titers for Opsonophagocytic Activity Against Vaccine Serotype 6C - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: as for outcome 36
Time Frame: as for outcome 6
Population: as for outcome 9
Arm/Group | 10PP-HD 2+1D Group | Synflorix 2+1D Group
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Concentrations of Antibodies Inhibiting Pneumococcal Pneumolysin Toxoid (Ply) Haemolysis Activity, or Hem-Ply Antibodies - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: The results of analysis of the anti-Ply haemolysis activity inhibition for Cohort 2 are not presented as assay was no longer available. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

39. Secondary Outcome: Concentrations of Antibodies Inhibiting Pneumococcal Pneumolysin Toxoid (Ply) Haemolysis Activity, or Hem-Ply Antibodies - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: The results of analysis of the anti-Ply haemolysis activity inhibition for Cohort 2 are not presented as assay was no longer available. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 9
Arm/Group | 10PP-HD 2+1D Group | Synflorix 2+1D Group
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Concentrations of Antibodies Against Diphtheria (Anti-D) and Tetanus (Anti-T) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule. Seroprotection rate = Anti-D or anti-T antibody concentrations ≥ 0.1 IU/mL.
Time Frame: At 1 month post-Dose 3 of the pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 99 | 99 | 98 | 99
IU/mL
  Anti-D 1 Mth post dose 3 | 2.499 [2.111 to 2.959] | 2.696 [2.381 to 3.053] | 2.874 [2.524 to 3.272] | 1.531 [1.330 to 1.762]
  Anti-T 1 Mth post dose 3 | 4.977 [4.127 to 6.002] | 5.113 [4.294 to 6.089] | 4.709 [3.994 to 5.551] | 4.047 [3.462 to 4.731]

41. Secondary Outcome: Concentrations of Antibodies Against Diphtheria (Anti-D) and Tetanus (Anti-T) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule. Seroprotection rate = Anti-D or anti-T antibody concentrations ≥ 0.1 IU/mL.
Time Frame: At 1 month post-Dose 2 of the pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 95 | 96
IU/mL
  Anti-D 1 Mth post dose 2 | 2.591 [2.213 to 3.033] | 2.560 [2.207 to 2.969]
  Anti-T 1 Mth post dose 2 | 5.714 [4.816 to 6.781] | 4.738 [3.905 to 5.749]

42. Secondary Outcome: Concentrations of Antibodies Against Bordetella Pertussis (Anti-BPT) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule. Seropositivity rate = Anti-BPT concentrations ≥ 15 EL.U/mL.
Time Frame: At 1 month post-Dose 3 of the pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 99 | 99 | 98 | 99
EL.U/mL | 111.9 [99.4 to 125.8] | 110.3 [99.3 to 122.5] | 105.8 [94.4 to 118.6] | 117.0 [105.0 to 130.3]

43. Secondary Outcome: Concentrations of Antibodies Against Bordetella Pertussis (Anti-BPT) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule. Seropositivity rate = Anti-BPT concentrations ≥ 15 EL.U/mL.
Time Frame: At 1 month post-Dose 2 of the pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 94 | 96
EL.U/mL | 123.2 [112.0 to 135.5] | 114.7 [101.3 to 129.9]

44. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl Ribitol Phosphate (Anti-PRP) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule. Seroprotection rate = Anti-PRP antibody concentrations ≥ 0.15 µg/mL.
Time Frame: At 1 month post-Dose 3 of the pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 99 | 99 | 98 | 99
µg/mL | 23.381 [19.326 to 28.287] | 19.397 [15.319 to 24.561] | 19.239 [15.085 to 24.537] | 18.981 [15.244 to 23.635]

45. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl Ribitol Phosphate (Anti-PRP) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule. Seroprotection rate = Anti-PRP antibody concentrations ≥ 0.15 µg/mL.
Time Frame: At 1 month post-Dose 2 of the pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 95 | 96
µg/mL | 21.274 [17.909 to 25.272] | 21.150 [17.427 to 25.669]

46. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B Surface Antigens (Anti-HBs) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule. Seroprotection rate = Anti-HB antibody concentrations ≥ 10 mIU/mL.
Time Frame: At 1 month post-Dose 3 of the pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 94 | 93 | 91 | 89
mIU/mL | 1235.8 [946.9 to 1612.9] | 1165.8 [910.7 to 1492.3] | 990.1 [757.6 to 1294.0] | 1206.6 [946.2 to 1538.7]

47. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B Surface Antigens (Anti-HBs) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule. Seroprotection rate = Anti-HB antibody concentrations ≥ 10 mIU/mL.
Time Frame: At 1 month post-Dose 2 of the pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 89 | 88
mIU/mL | 1318.5 [1062.5 to 1636.3] | 976.5 [724.2 to 1316.8]

48. Secondary Outcome: Antibody Titers Against Poliovirus 1, 2 and 3 (Anti-Polio, Anti-Polio 2 and Anti-Polio 3) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule. Seroprotection rate = Anti-Polio titers ≥ 8.
Time Frame: At 1 month post-Dose 3 of the pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 97 | 92 | 91 | 94
Titers
  Anti-Polio 1 - 1 Mth post dose 3 | 413.2 [287.0 to 594.9] | 314.8 [202.7 to 488.7] | 447.9 [278.5 to 720.1] | 398.3 [256.6 to 618.3]
  Anti-Polio 2 - 1 Mth post dose 3: number analyzed (Participants) | 76 | 78 | 76 | 73
  Anti-Polio 2 - 1 Mth post dose 3 | 545.8 [371.6 to 801.6] | 619.5 [462.0 to 830.7] | 514.2 [353.8 to 747.2] | 536.9 [400.6 to 719.6]
  Anti-Polio 3 - 1 Mth post dose 3: number analyzed (Participants) | 80 | 88 | 82 | 84
  Anti-Polio 3 - 1 Mth post dose 3 | 135.4 [91.5 to 200.5] | 166.0 [124.5 to 221.5] | 110.1 [72.5 to 167.2] | 191.8 [129.4 to 284.4]

49. Secondary Outcome: Antibody Titers Against Poliovirus 1, 2 and 3 (Anti-Polio, Anti-Polio 2 and Anti-Polio 3) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule. Seroprotection rate = Anti-Polio titers ≥ 8.
Time Frame: At 1 month post-Dose 2 of the pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 87 | 93
Titers
  Anti-Polio 1 - 1 Mth post dose 2 | 330.3 [208.6 to 523.0] | 415.6 [286.7 to 602.6]
  Anti-Polio 2 - 1 Mth post dose 2: number analyzed (Participants) | 75 | 82
  Anti-Polio 2 - 1 Mth post dose 2 | 486.7 [319.7 to 741.1] | 702.9 [529.6 to 932.8]
  Anti-Polio 3 - 1 Mth post dose 2: number analyzed (Participants) | 75 | 80
  Anti-Polio 3 - 1 Mth post dose 2 | 106.9 [71.8 to 159.1] | 181.1 [131.7 to 249.0]

50. Secondary Outcome: Concentrations of Antibodies Against Measles (Anti-Measles) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule. Seroprotection rate = Anti-Measles antibody concentrations ≥ 150 mIU/mL.
Time Frame: At 3 months (Mth) post-vaccination with Stamaril™/M-Vac™
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 90 | 95 | 96 | 86
mIU/mL | 329.2 [272.6 to 397.5] | 298.6 [254.9 to 349.8] | 295.8 [237.2 to 368.8] | 274.1 [227.7 to 330.0]

51. Secondary Outcome: Concentrations of Antibodies Against Measles (Anti-Measles) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule. Seroprotection rate = Anti-Measles antibody concentrations ≥ 150 mIU/mL.
Time Frame: At 3 months (Mth) post-vaccination with Stamaril™/M-Vac™
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 96 | 94
mIU/mL | 284.5 [240.9 to 336.0] | 305.9 [256.5 to 364.8]

52. Secondary Outcome: Titers of Antibodies Against Yellow Fever (Anti-YF) - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule. Seroprotection rate = Anti-yellow fever antibody titers ≥ 10.
Time Frame: At 3 months (Mth) post-vaccination with Stamaril™/M-Vac™
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 97 | 95 | 97 | 98
Titers | 334.0 [250.6 to 445.1] | 264.7 [201.0 to 348.5] | 379.9 [293.2 to 492.2] | 306.7 [242.9 to 387.3]

53. Secondary Outcome: Titers of Antibodies Against Yellow Fever (Anti-YF) - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule. Seroprotection rate = Anti-yellow fever antibody titers ≥ 10.
Time Frame: At 3 months (Mth) post-vaccination with Stamaril™/M-Vac™
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 94 | 95
Titers | 342.0 [252.2 to 463.7] | 239.0 [176.0 to 324.5]

54. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - For Cohort2/Step 2 Subjects Receiving the 3+0 Schedule.
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm). This outcome concerns Cohort2/Step 2 subjects receiving the 3+0 Schedule.
Time Frame: Within the 4-day (Days 0-3) periods post vaccination with 3 doses of pneumococcal vaccine (10PP vaccine, Synflorix™ or Prevnar 13™), across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Prevnar 13 3+0d Group: This group consisted in infants aged 8-10 weeks at first vaccination enrolled as part the Cohort 2/Step 2 of the study who received 3 doses of Prevnar 13™ and EPI vaccines according to a 3+0 Schedule. That is, subjects received 3 doses of Prevnar 13™, co-administered with Tritanrix™-HepB/Hib and Polio Sabin™ at 2-3-4 months of age (Day 0, Month 1 and Month 2), followed by one dose of each of the M-Vac™, Stamaril™ and Polio Sabin™ vaccines administered at approximately 9 months of age. Prevnar 13™ was administered intramuscularly into the right thigh; Tritanrix™-HepB/Hib, M-Vac™ and Stamaril™ were administered intramuscularly into the left thigh; Polio Sabin™ was administered orally.
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar 13 3+0d Group
Number analyzed (Participants) | 200 | 200 | 200 | 200
Participants
  Any pain | 108 | 121 | 123 | 115
  Grade 3 pain | 0 | 1 | 0 | 0
  Any redness | 8 | 7 | 9 | 5
  Grade 3 redness | 0 | 1 | 1 | 0
  Any swelling | 30 | 45 | 40 | 37
  Grade 3 swelling | 7 | 10 | 17 | 7

55. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - For Cohort2/Step 2 Subjects Receiving the 2+1 Schedule.
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm). This outcome concerns Cohort2/Step 2 subjects receiving the 2+1 Schedule.
Time Frame: Within the 4-day (Days 0-3) periods post vaccination with the 2 first doses of pneumococcal vaccine (10PP vaccine or Synflorix™), across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 200 | 200
Participants
  Any pain | 97 | 102
  Grade 3 pain | 1 | 1
  Any redness | 3 | 5
  Grade 3 redness | 0 | 0
  Any swelling | 35 | 31
  Grade 3 swelling | 9 | 4

56. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - For Cohort2/Step 2 Subjects Receiving the 2+1 Schedule.
Description: as for outcome 55
Time Frame: Within the 4-day (Days 0-3) period post vaccination with Dose 3 of pneumococcal vaccine (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 191 | 195
Participants
  Any pain | 21 | 26
  Grade 3 pain | 0 | 0
  Any redness | 0 | 0
  Grade 3 redness | 0 | 0
  Any swelling | 4 | 8
  Grade 3 swelling | 1 | 3

57. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination - For Step 2/Cohort 2 Subjects Receiving the 3+0 Schedule
Description: Assessed solicited general symptoms were Drowsiness, Fever (axillary temperature higher than [≥] 37.5 degrees Celsius [°C]), Irritability/Fussiness and Loss of appetite. Any = Occurrence of the specified solicited general symptom, regardless of intensity. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Fever = Axillary temperature higher than (>) 39.5°C. Grade 3 Irritability/fussiness = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. This outcome concerns Step 2/Cohort 2 subjects receiving the 3+0 Schedule.
Time Frame: as for outcome 54
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar 13 3+0d Group
Number analyzed (Participants) | 200 | 200 | 200 | 200
Participants
  Any Drowsiness | 43 | 46 | 38 | 44
  Grade 3 Drowsiness | 0 | 0 | 0 | 0
  Related Drowsiness | 43 | 45 | 38 | 43
  Any Irritability/fussiness | 139 | 133 | 141 | 136
  Grade 3 Irritability/fussiness | 6 | 4 | 4 | 7
  Related Irritability/fussiness | 138 | 132 | 138 | 136
  Any Loss of appetite | 32 | 30 | 27 | 34
  Grade 3 Loss of appetite | 0 | 0 | 1 | 0
  Related Loss of appetite | 32 | 29 | 26 | 34
  Any Fever | 104 | 100 | 105 | 106
  Grade 3 Fever | 0 | 0 | 0 | 0
  Related Fever | 102 | 100 | 104 | 104

58. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination - For Step 2/Cohort 2 Subjects Receiving the 2+1 Schedule
Description: Assessed solicited general symptoms were Drowsiness, Fever (axillary temperature higher than [≥] 37.5 degrees Celsius [°C]), Irritability/Fussiness and Loss of appetite. Any = Occurrence of the specified solicited general symptom, regardless of intensity. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Fever = Axillary temperature higher than (>) 39.5°C. Grade 3 Irritability/fussiness = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. This outcome concerns Step 2/Cohort 2 subjects receiving the 2+1 Schedule.
Time Frame: as for outcome 55
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 200 | 200
Participants
  Any Drowsiness | 47 | 44
  Grade 3 Drowsiness | 0 | 0
  Related Drowsiness | 46 | 43
  Any Fever | 92 | 84
  Grade 3 Fever | 0 | 0
  Related Fever | 89 | 84
  Any Irritability/fussiness | 131 | 128
  Grade 3 Irritability/fussiness | 1 | 2
  Related Irritability/fussiness | 128 | 126
  Any Loss of appetite | 24 | 25
  Grade 3 Loss of appetite | 0 | 0
  Related Loss of appetite | 24 | 24

59. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination - For Step 2/Cohort 2 Subjects Receiving the 2+1 Schedule
Description: as for outcome 58
Time Frame: Within the 4-day (Days 0-3) period post vaccination with Dose 3 of pneumococcal vaccine (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 191 | 195
Participants
  Any Drowsiness | 12 | 4
  Grade 3 Drowsiness | 0 | 0
  Related Drowsiness | 12 | 4
  Any Fever | 32 | 27
  Grade 3 Fever | 0 | 1
  Related Fever | 30 | 25
  Any Irritability/fussiness | 27 | 19
  Grade 3 Irritability/fussiness | 0 | 0
  Related Irritability/fussiness | 27 | 19
  Any Loss of appetite | 3 | 5
  Grade 3 Loss of appetite | 0 | 0
  Related Loss of appetite | 3 | 4

60. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - For Step 2/Cohort 2 Subjects Receiving the 3+0 Schedule
Description: An unsolicited AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination. This outcome concerns Step 2/Cohort 2 subjects receiving the 3+0 Schedule.
Time Frame: Within the 31-day (Days 0-30) periods post vaccination with 3 doses of pneumococcal vaccine (10PP vaccine, Synflorix™ or Prevnar 13™), across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar 13 3+0d Group
Number analyzed (Participants) | 200 | 200 | 200 | 200
Participants | 113 | 114 | 123 | 114

61. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - For Step 2/Cohort 2 Subjects Receiving the 2+1 Schedule
Description: An unsolicited AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination. This outcome concerns Step 2/Cohort 2 subjects receiving the 2+1 Schedule.
Time Frame: Within the 31-day (Days 0-30) periods post vaccination with the first 2 doses of pneumococcal vaccine (10PP vaccine or Synflorix™), across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 200 | 200
Participants | 84 | 95

62. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - For Step 2/Cohort 2 Subjects Receiving the 2+1 Schedule
Description: as for outcome 61
Time Frame: Within the 31-day (Days 0-30) period post vaccination with Dose 3 of pneumococcal vaccine (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 191 | 195
Participants | 7 | 2

63. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) - For Step 2/Cohort 2 Subjects Receiving the 3+0 Schedule
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity. These should also be considered serious: invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation. Any = Occurrence of an SAE, regardless of relationship to vaccination. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: From Day 0 to Month 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 200 | 200 | 200 | 200
Participants | 1 | 4 | 3 | 2

64. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) - For Step 2/Cohort 2 Subjects Receiving the 2+1 Schedule
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity. These should also be considered serious: invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation. Any = Occurrence of an SAE, regardless of relationship to vaccination. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: From Day 0 to Month 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 200 | 200
Participants | 4 | 5

65. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (Any) in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: Numbers of subjects with positive nasopharyngeal sample were calculated per group, at each swab time point. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 165 | 158 | 166 | 155
  At 5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 194 | 193
  At 5 Mth post dose 3 | 166 | 161 | 176 | 168
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 191
  At 8 Mth post dose 3 | 174 | 166 | 174 | 171

66. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (Any) in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: Numbers of subjects with positive nasopharyngeal sample were calculated per group, at each swab time point. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 159 | 162
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 194
  At 5 Mth post-dose 2 | 164 | 173
  At 3 Mth post-dose 3: number analyzed (Participants) | 190 | 193
  At 3 Mth post-dose 3 | 178 | 176

67. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (10Pn-PD-DiT Vaccine Serotypes) in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: Numbers of subjects with positive nasopharyngeal sample were calculated per group, at each swab time point. A Streptococcus. Pneumoniae (S. pn). vaccine pneumococcal serotype was defined as any of the pneumococcal S. pn. vaccine serotypes, e. a. serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 24 | 31 | 34 | 29
  At 5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 194 | 193
  At 5 Mth post dose 3 | 25 | 23 | 28 | 30
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 191
  At 8 Mth post dose 3 | 24 | 15 | 16 | 21

68. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (10Pn-PD-DiT Vaccine Serotypes) in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: Numbers of subjects with positive nasopharyngeal sample were calculated per group, at each swab time point. A Streptococcus. Pneumoniae (S. pn). vaccine pneumococcal serotype was defined as any of the pneumococcal S. pn. vaccine serotypes, e. a. serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 27 | 24
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 194
  At 5 Mth post-dose 2 | 24 | 23
  At 3 Mth post-dose 3: number analyzed (Participants) | 190 | 193
  At 3 Mth post-dose 3 | 18 | 19

69. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (Synflorix Related Serotypes) in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: Related serotype = any serotype belonging to the same serogroup as the Synflorix vaccine serotypes, but different from the vaccine serotypes, was considered for the analyses of carriage of S. pneumoniae cross-related serotypes. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 57 | 56 | 60 | 48
  At 5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 194 | 193
  At 5 Mth post dose 3 | 54 | 48 | 58 | 46
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 191
  At 8 Mth post dose 3 | 45 | 42 | 47 | 42

70. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae (Synflorix Related Serotypes) in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: Related serotype = any serotype belonging to the same serogroup as the Synflorix vaccine serotypes, but different from the vaccine serotypes, was considered for the analyses of carriage of S. pneumoniae cross-related serotypes. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 62 | 50
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 194
  At 5 Mth post-dose 2 | 45 | 49
  At 3 Mth post-dose 3: number analyzed (Participants) | 190 | 193
  At 3 Mth post-dose 3 | 58 | 52

71. Secondary Outcome: Number of Subjects With Haemophilus Influenzae in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 195 | 196
Participants
  At 1 Mth post dose 3: number analyzed (Participants) | 192 | 194 | 195 | 196
  At 1 Mth post dose 3 | 29 | 33 | 28 | 37
  At 5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 193 | 193
  At 5 Mth post dose 3 | 27 | 28 | 28 | 30
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 191
  At 8 Mth post dose 3 | 9 | 13 | 12 | 9

72. Secondary Outcome: Number of Subjects With Haemophilus Influenzae in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 26 | 23
  At 5 Mth post-dose 2: number analyzed (Participants) | 187 | 194
  At 5 Mth post-dose 2 | 20 | 32
  At 3 Mth post-dose 3: number analyzed (Participants) | 190 | 193
  At 3 Mth post-dose 3 | 9 | 11

73. Secondary Outcome: Number of Subjects With Moraxella Catarrhalis in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: Positive cultures of other bacterial pathogens [such as S. aureus, Streptococcus pyogenes (Group A streptococci) and Moraxella catarrhalis] identified in the nasopharynx were analyzed. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 88 | 98 | 104 | 100
  At 5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 194 | 193
  At 5 Mth post dose 3 | 72 | 73 | 78 | 88
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 191
  At 8 Mth post dose 3 | 74 | 67 | 70 | 74

74. Secondary Outcome: Number of Subjects With Moraxella Catarrhalis in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: Positive cultures of other bacterial pathogens [such as S. aureus, Streptococcus pyogenes (Group A streptococci) and Moraxella catarrhalis] identified in the nasopharynx were analyzed. This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 86 | 93
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 194
  At 5 Mth post-dose 2 | 73 | 84
  At 3 Mth post-dose 3: number analyzed (Participants) | 190 | 193
  At 3 Mth post-dose 3 | 56 | 83

75. Secondary Outcome: Number of Subjects With Group A Streptococcus in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: Positive cultures of other bacterial pathogens [such as S. aureus, Streptococcus pyogenes (Group A streptococci) and Moraxella catarrhalis] identified in the nasopharynx were analyzed.This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 5 | 4 | 5 | 4
  At 5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 194 | 193
  At 5 Mth post dose 3 | 4 | 3 | 4 | 1
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 191
  At 8 Mth post dose 3 | 4 | 6 | 7 | 6

76. Secondary Outcome: Number of Subjects With Group A Streptococcus in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: as for outcome 74
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 6 | 4
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 194
  At 5 Mth post-dose 2 | 2 | 4
  At 3 Mth post-dose 3: number analyzed (Participants) | 190 | 193
  At 3 Mth post-dose 3 | 5 | 2

77. Secondary Outcome: Number of Subjects With Staphylococcus Aureus in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: as for outcome 73
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine, Synflorix™ or Prevnar 13™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 44 | 44 | 54 | 50
  At 5 Mth post dose 3: number analyzed (Participants) | 193 | 192 | 194 | 193
  At 5 Mth post dose 3 | 36 | 37 | 39 | 37
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 194 | 191
  At 8 Mth post dose 3 | 13 | 17 | 25 | 11

78. Secondary Outcome: Number of Subjects With Staphylococcus Aureus in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: as for outcome 74
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 46 | 62
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 194
  At 5 Mth post-dose 2 | 32 | 40
  At 3 Mth post-dose 3: number analyzed (Participants) | 190 | 193
  At 3 Mth post-dose 3 | 21 | 17

79. Secondary Outcome: Number of Subjects With Acquisition of Non-vaccine Serotypes/Serogroups of Streptococcus Pneumoniae in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 124 | 106 | 120 | 112
  At 5 Mth post dose 3: number analyzed (Participants) | 192 | 191 | 194 | 191
  At 5 Mth post dose 3 | 108 | 122 | 131 | 126
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 193 | 190
  At 8 Mth post dose 3 | 121 | 115 | 122 | 122

80. Secondary Outcome: Number of Subjects With Acquisition of Non-vaccine Serotypes/Serogroups of Streptococcus Pneumoniae in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 117 | 128
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 193
  At 5 Mth post-dose 2 | 119 | 138
  At 3 Mth post-dose 3: number analyzed (Participants) | 188 | 192
  At 3 Mth post-dose 3 | 129 | 117

81. Secondary Outcome: Number of Subjects With Acquisition of Any New Streptococcus Pneumoniae in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 136 | 130 | 142 | 133
  At 5 Mth post dose 3: number analyzed (Participants) | 192 | 191 | 194 | 191
  At 5 Mth post dose 3 | 128 | 130 | 145 | 142
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 193 | 190
  At 8 Mth post dose 3 | 139 | 128 | 136 | 135

82. Secondary Outcome: Number of Subjects With Acquisition of Any New Streptococcus Pneumoniae in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 136 | 141
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 193
  At 5 Mth post-dose 2 | 136 | 155
  At 3 Mth post-dose 3: number analyzed (Participants) | 188 | 192
  At 3 Mth post-dose 3 | 144 | 131

83. Secondary Outcome: Number of Subjects With Acquisition of Haemophilus Influenzae Strains Identified With Polymerase Chain Reaction Differentiation in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 3+0 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 3+0 Schedule.
Time Frame: At 1, 5 and 8 months (Mth) post-Dose 3 of pneumococcal vaccine administered (10PP vaccine or Synflorix™)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 3+0d Group | 10PP-LD 3+0d Group | Synflorix 3+0d Group | Prevnar13 3+0d Group
Number analyzed (Participants) | 193 | 194 | 196 | 196
Participants
  At 1 Mth post dose 3 | 17 | 21 | 16 | 19
  At 5 Mth post dose 3: number analyzed (Participants) | 192 | 191 | 194 | 191
  At 5 Mth post dose 3 | 24 | 23 | 25 | 24
  At 8 Mth post dose 3: number analyzed (Participants) | 189 | 189 | 193 | 190
  At 8 Mth post dose 3 | 9 | 10 | 10 | 6

84. Secondary Outcome: Number of Subjects With Acquisition of Haemophilus Influenzae Strains Identified With Polymerase Chain Reaction Differentiation in the Nasopharynx - For Cohort 2/Step 2 Subjects Receiving the 2+1 Schedule
Description: This outcome concerns subjects enrolled in Cohort 2/Step 2 receiving the 2+1 Schedule.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 197 | 197
Participants
  At 1 Mth post-dose 2 | 12 | 12
  At 5 Mth post-dose 2: number analyzed (Participants) | 189 | 193
  At 5 Mth post-dose 2 | 20 | 25
  At 3 Mth post-dose 3: number analyzed (Participants) | 188 | 192
  At 3 Mth post-dose 3 | 9 | 8

85. Other Pre Specified Outcome: Description of Non-Vaccine-Type S.Pneumoniae Samples Isolated From Nasopharyngeal Swabs Before and After Vaccination for the Ply Gene - Cohort 2
Description: Isolates from the Prev13_3D group were not selected. Samples were distributed evenly in the 5 groups and across time points: 10 isolates from pre-vaccination, 20 at Month 3, 20 at Month 7 and 20 at Month 10. Only samples displaying non-vaccine and non-vaccine related serotypes (all serotypes except serotypes 1, 4, 5 and 14 and serotypes belonging to the serogroups 6, 7, 9, 18, 19 and 23) were selected in systematic (equal number across groups) but non-random manner. Samples were described as follows: samples with gene detected (Positive isolates) with sequenced protein, number of protein Variants, number of isolates with Variant 1 (100% identity with vaccine sequence).
Time Frame: At Month 0 (Pre-vaccination), Month 3 (1 month [m] post-dose [P] III-3+0 schedule or PII-2+1 schedule), Month 7 (5 m PIII - 3+0 schedule or PII-2+1 schedule) or at Month 10 (8 m PIII - 3+0 schedule or 3 m post-booster-2+1 schedule)
Population: The analysis was performed on vaccinated subjects with at least one vaccine administration documented for which S. pneumoniae isolates samples were selected for ply and phtD gene sequencing.
Measure: Number; unit: Samples
Groups:
- Total "All 5" Group: A subset of samples selected for ply and phtD gene sequencing of S. pneumoniae isolates, isolated from nasopharyngeal samples across all time points and across study groups of Cohort 2 (Prev13_3 group was excluded).
Arm/Group | Total "All 5" Group
Number analyzed (Participants) | 350
Samples
  Positive isolates | 347
  Protein sequenced | 347
  Protein variants | 18
  Samples with Variant 1 | 216

86. Other Pre Specified Outcome: Description of Non-Vaccine-Type S.Pneumoniae Samples Isolated From Nasopharyngeal Swabs Before and After Vaccination for the PhtD Gene - Cohort 2
Description: as for outcome 85
Time Frame: as for outcome 85
Population: as for outcome 85
Measure: Number; unit: Samples
Arm/Group | Total "All 5" Group
Number analyzed (Participants) | 350
Samples
  Positive isolates | 342
  Protein sequenced | 321
  Protein variants | 84
  Samples with Variant 1 | 1

87. Other Pre Specified Outcome: Number of Samples With Ply Protein Variants Classified by Number of Amino Acids (AA) Mutation Versus Vaccine Sequence in a Subset of Non-Vaccine-Type S.Pneumoniae Isolates From Nasopharyngeal Swabs - Cohort 2
Description: Overall, 18 different Ply protein sequences were identified: 5 protein variants previously described (e.g. variants 1, 2, 7, 11 and 15), plus 13 new protein variants which are referred to as variants GSK21 to GSK33. The number of Amino Acids (AA) mutation versus vaccine sequence has been specified for each Ply variant. The samples without gene detected were considered as negative for Ply (Ply negative).
Time Frame: At Month 0 (Pre-vaccination), Month 3 (1 month [m] post-dose [P] III-3+0 schedule or PII-2+1 schedule), Month 7 (5 m PIII - 3+0 schedule or PII-2+1 schedule) and Month 10 (8 m PIII - 3+0 schedule or 3 m post-booster-2+1 schedule)
Population: as for outcome 85
Measure: Number; unit: Samples
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Samples
  Variant 1 - AA = 0 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant 1 - AA = 0 at Month 0 | 5 | 8 | 7 | 4 | 8
  Variant 2 - AA = 1 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant 2 - AA = 1 at Month 0 | 4 | 0 | 1 | 4 | 1
  Variant 15 - AA = 1 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant 15 - AA = 1 at Month 0 | 1 | 0 | 0 | 2 | 0
  Variant GSK 24 - AA = 1 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant GSK 24 - AA = 1 at Month 0 | 0 | 0 | 1 | 0 | 0
  Variant GSK 28 - AA = 1 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant GSK 28 - AA = 1 at Month 0 | 0 | 0 | 1 | 0 | 0
  Variant GSK 33 - AA = 3 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant GSK 33 - AA = 3 at Month 0 | 0 | 0 | 0 | 0 | 1
  Variant GSK 30 - AA = 4 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant GSK 30 - AA = 4 at Month 0 | 0 | 1 | 0 | 0 | 0
  Variant GSK 31 - AA = 6 at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variant GSK 31 - AA = 6 at Month 0 | 0 | 1 | 0 | 0 | 0
  Ply negative at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Ply negative at Month 0 | 0 | 0 | 0 | 0 | 0
  Variant 1 - AA = 0 at Month 3 | 11 | 13 | 10 | 14 | 9
  Variant 2 - AA = 1 at Month 3 | 4 | 7 | 6 | 4 | 8
  Variant 15 - AA = 1 at Month 3 | 2 | 0 | 2 | 1 | 0
  Variant GSK 24 - AA = 1 at Month 3 | 2 | 0 | 1 | 1 | 0
  Variant 11 - AA = 2 at Month 3 | 0 | 0 | 0 | 0 | 1
  Variant GSK 23 - AA = 2 at Month 3 | 0 | 0 | 0 | 0 | 2
  Ply negative at Month 3 | 1 | 0 | 1 | 0 | 0
  Variant 1 - AA = 0 at Month 7 | 14 | 15 | 10 | 13 | 10
  Variant 2 - AA = 1 at Month 7 | 4 | 4 | 6 | 4 | 7
  Variant 15 - AA = 1 at Month 7 | 2 | 0 | 1 | 1 | 1
  Variant GSK 24 - AA = 1 at Month 7 | 0 | 0 | 0 | 1 | 0
  Variant GSK 29 - AA = 1 at Month 7 | 0 | 0 | 0 | 0 | 1
  Variant 7 - AA = 2 at Month 7 | 0 | 1 | 1 | 1 | 0
  Variant GSK 21 - AA = 2 at Month 7 | 0 | 0 | 1 | 0 | 0
  Variant GSK 23 - AA = 2 at Month 7 | 0 | 0 | 0 | 0 | 1
  Variant GSK 27 - AA = 2 at Month 7 | 0 | 0 | 1 | 0 | 0
  Ply negative at Month 7 | 0 | 0 | 0 | 0 | 0
  Variant 1 - AA = 0 at Month 10 | 12 | 15 | 12 | 12 | 14
  Variant 2 - AA = 1 at Month 10 | 5 | 2 | 6 | 5 | 4
  Variant 15 - AA = 1 at Month 10 | 1 | 1 | 0 | 2 | 1
  Variant GSK 24 - AA = 1 at Month 10 | 0 | 0 | 0 | 0 | 1
  Variant GSK 25 - AA = 1 at Month 10 | 0 | 1 | 0 | 0 | 0
  Variant 7 - AA = 2 at Month 10 | 1 | 0 | 0 | 1 | 0
  Variant GSK 22 - AA = 2 at Month 10 | 0 | 0 | 1 | 0 | 0
  Variant GSK 26 - AA = 4 at Month 10 | 0 | 0 | 1 | 0 | 0
  Variant GSK 32 - AA = 7 at Month 10 | 1 | 0 | 0 | 0 | 0
  Ply negative at Month 10 | 0 | 1 | 0 | 0 | 0

88. Other Pre Specified Outcome: Percentage (Median and Mean) of Protein Identity Relative to Amino Acid Sequence of Ply Protein in the Vaccine for a Subset of Non-Vaccine-Type S.Pneumoniae Isolates From Nasopharyngeal Swabs - Cohort 2
Description: Protein sequence identity was compared to vaccine sequence. Mean and median was calculated and expressed as percentage.
Time Frame: as for outcome 87
Population: as for outcome 85
Measure: Number; unit: Percentage of protein identity
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Percentage of protein identity
  Median at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Median at Month 0 | 99.90 | 100 | 100 | 99.79 | 100
  Mean at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Mean at Month 0 | 99.90 | 99.79 | 99.94 | 99.87 | 99.92
  Median at Month 3: number analyzed (Participants) | 19 | 20 | 19 | 20 | 20
  Median at Month 3 | 100 | 100 | 100 | 100 | 99.79
  Mean at Month 3: number analyzed (Participants) | 19 | 20 | 19 | 20 | 20
  Mean at Month 3 | 99.91 | 99.93 | 99.90 | 99.94 | 99.85
  Median at Month 7 | 100 | 100 | 99.90 | 100 | 99.90
  Mean at Month 7 | 99.94 | 99.94 | 99.86 | 99.92 | 99.88
  Median at Month 10: number analyzed (Participants) | 20 | 19 | 20 | 20 | 20
  Median at Month 10 | 100 | 100 | 100 | 100 | 100
  Mean at Month 10: number analyzed (Participants) | 20 | 19 | 20 | 20 | 20
  Mean at Month 10 | 99.84 | 99.95 | 99.87 | 99.91 | 99.94

89. Other Pre Specified Outcome: Number of Samples With PhtD Protein Variants in a Subset of Non-Vaccine-Type S.Pneumoniae Isolates From Nasopharyngeal Swabs - Cohort 2
Description: Because of high variants heterogeneity in each group (no major variant), the impact of vaccination on variant prevalence was not analysed. PhtD sequences were detected in some samples but no consensus sequence could be obtained they were defined as mixed sequences (Mix). The samples without gene detected were considered as negative for PhtD (PhtD negative).
Time Frame: as for outcome 87
Population: as for outcome 85
Measure: Number; unit: Samples
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Samples
  Variants number at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Variants number at Month 0 | 10 | 6 | 9 | 9 | 7
  Mix number at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  Mix number at Month 0 | 0 | 1 | 1 | 0 | 2
  PhtD negative at Month 0: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
  PhtD negative at Month 0 | 0 | 2 | 0 | 1 | 1
  Variants number at Month 3 | 16 | 16 | 18 | 16 | 16
  Mix number at Month 3 | 1 | 1 | 0 | 3 | 1
  PhtD negative at Month 3 | 1 | 0 | 1 | 0 | 0
  Variants number at Month 7 | 13 | 14 | 17 | 13 | 12
  Mix number at Month 7 | 0 | 2 | 1 | 1 | 1
  PhtD negative at Month 7 | 0 | 0 | 0 | 0 | 0
  Variants number at Month 10 | 13 | 12 | 13 | 15 | 11
  Mix number at Month 10 | 1 | 0 | 1 | 1 | 3
  PhtD negative at Month 10 | 1 | 1 | 0 | 0 | 0

90. Other Pre Specified Outcome: Percentage (Median and Mean) of Protein Identity Relative to Amino Acid Sequence of PhtD Protein in the Vaccine for a Subset of Non-Vaccine-Type S.Pneumoniae Isolates From Nasopharyngeal Swabs - Cohort 2
Description: Protein sequence identity was compared to vaccine sequence. Mean and median was calculated and expressed as percentage.
Time Frame: as for outcome 87
Population: as for outcome 85
Measure: Number; unit: Percentage of protein identity
Arm/Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
Number analyzed (Participants) | 20 | 19 | 19 | 19 | 19
Percentage of protein identity
  Median at Month 0: number analyzed (Participants) | 10 | 7 | 9 | 9 | 7
  Median at Month 0 | 96.3 | 96.7 | 95.8 | 96.7 | 95.7
  Mean at Month 0: number analyzed (Participants) | 10 | 7 | 9 | 9 | 7
  Mean at Month 0 | 95.2 | 97.0 | 96.7 | 96.3 | 96.3
  Median at Month 3: number analyzed (Participants) | 18 | 19 | 19 | 17 | 19
  Median at Month 3 | 96.6 | 97.7 | 96.6 | 96.3 | 95.7
  Mean at Month 3: number analyzed (Participants) | 18 | 19 | 19 | 17 | 19
  Mean at Month 3 | 96.4 | 97.4 | 96.2 | 94.6 | 93.1
  Median at Month 7: number analyzed (Participants) | 20 | 18 | 19 | 19 | 19
  Median at Month 7 | 97.6 | 96.2 | 97.4 | 97.6 | 95.7
  Mean at Month 7: number analyzed (Participants) | 20 | 18 | 19 | 19 | 19
  Mean at Month 7 | 96.7 | 95.6 | 95.7 | 96.7 | 94.7
  Median at Month 10: number analyzed (Participants) | 18 | 19 | 19 | 19 | 17
  Median at Month 10 | 97.2 | 97.6 | 96.8 | 96.9 | 97.6
  Mean at Month 10: number analyzed (Participants) | 18 | 19 | 19 | 19 | 17
  Mean at Month 10 | 95.5 | 97.3 | 94.1 | 95.4 | 94.9

ADVERSE EVENTS:
Time Frame: Solicited symptoms during the 4-day post-vaccination period in Cohort 1 and 2. Unsolicited AEs during 31-day post-vaccination period in Cohort 1 and 2. SAEs from Month 0 to Month 6 in Cohort 1 and from Month 0 to Month 10 in Cohort 2.
Arm/Group | 10PP-HD 1d Group | Prevnar 13 1d Group | 10PP-LD 3+0d Group | 10PP-HD 3+0d Group | Synflorix 3+0d Group | Prevnar 13 3+0d Group | 10PP-HD 2+1d Group | Synflorix 2+1d Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/200 | 1/200 | 0/200 | 2/200 | 2/200 | 1/200
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 1/200 | 4/200 | 3/200 | 2/200 | 4/200 | 5/200
Other Adverse Events (participants affected / at risk) | 9/60 | 3/60 | 186/200 | 191/200 | 193/200 | 188/200 | 189/200 | 184/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10PP-HD 1d Group (N=60) | Prevnar 13 1d Group (N=60) | 10PP-LD 3+0d Group (N=200) | 10PP-HD 3+0d Group (N=200) | Synflorix 3+0d Group (N=200) | Prevnar 13 3+0d Group (N=200) | 10PP-HD 2+1d Group (N=200) | Synflorix 2+1d Group (N=200)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 10PP-HD 1d Group (N=60) | Prevnar 13 1d Group (N=60) | 10PP-LD 3+0d Group (N=200) | 10PP-HD 3+0d Group (N=200) | Synflorix 3+0d Group (N=200) | Prevnar 13 3+0d Group (N=200) | 10PP-HD 2+1d Group (N=200) | Synflorix 2+1d Group (N=200)
Fever (axillary temperature ≥ 37.5°C) (General disorders) | 4 | 2 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Solicited general symptom reported during the 4-day post-vaccination period in Cohort 1
Pain (General disorders) | 0/0 | 0/0 | 108 | 121 | 123 | 115 | 0/0 | 0/0 — Solicited local symptom reported during the 4-day post-vaccination periods, across doses - in Cohort 2 3+0 Schedule subjects
Swelling (General disorders) | 0/0 | 0/0 | 30 | 45 | 40 | 37 | 0/0 | 0/0 — Solicited local symptom reported during the 4-day post-vaccination periods, across doses - in Cohort 2 3+0 Schedule subjects
Pain (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 97 | 102 — Solicited local symptom reported during the 4-day periods after vaccination with Doses 1 and 2, across doses - in Cohort 2 2+1 Schedule subjects
Swelling (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 35 | 31 — Solicited local symptom reported during the 4-day periods after vaccination with Doses 1 and 2, across doses - in Cohort 2 2+1 Schedule subjects
Pain (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 21/191 | 26/195 — Solicited local symptom reported during the 4-day period after vaccination with Dose 3 - in Cohort 2 2+1 Schedule subjects
Somnolence (Nervous system disorders) | 0/0 | 0/0 | 43 | 46 | 38 | 44 | 0/0 | 0/0 — Solicited general symptom reported during the 4-day post-vaccination periods, across doses - in Cohort 2 3+0 Schedule subjects
Irritability (Psychiatric disorders) | 0/0 | 0/0 | 139 | 133 | 141 | 136 | 0/0 | 0/0 — Solicited general symptom reported during the 4-day post-vaccination periods, across doses - in Cohort 2 3+0 Schedule subjects
Decreased appetite (Metabolism and nutrition disorders) | 0/0 | 0/0 | 32 | 30 | 27 | 34 | 0/0 | 0/0 — Solicited general symptom reported during the 4-day post-vaccination period, across doses - in Cohort 2 3+0 Schedule subjects
Pyrexia (General disorders) | 0/0 | 0/0 | 105 | 104 | 106 | 106 | 0/0 | 0/0 — Solicited general symptom reported during the 4-day post-vaccination period, across doses - in Cohort 2 3+0 Schedule subjects
Somnolence (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 47 | 44 — Solicited general symptom reported during the 4-day periods after vaccination with Doses 1 and 2, across doses - in Cohort 2 2+1 Schedule subjects
Irritability (Psychiatric disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 131 | 128 — Solicited general symptom reported during the 4-day periods after vaccination with Doses 1 and 2, across doses - in Cohort 2 2+1 Schedule subjects
Decreased appetite (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 24 | 25 — Solicited general symptom reported during the 4-day periods after vaccination with Doses 1 and 2, across doses - in Cohort 2 2+1 Schedule subjects
Pyrexia (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 93 | 89 — Solicited general symptom reported during the 4-day periods after vaccination with Doses 1 and 2, across doses - in Cohort 2 2+1 Schedule subjects
Somnolence (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 12/191 | 4/195 — Solicited general symptom reported during the 4-day period after vaccination with Dose 3 - in Cohort 2 2+1 Schedule subjects
Irritability (Psychiatric disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 27/191 | 19/195 — Solicited general symptom during the 4-day period after vaccination with Dose 3 - in Cohort 2 2+1 Schedule subjects
Pyrexia (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 32/191 | 27/195 — Solicited general symptom reported during the 4-day period after vaccination with Dose 3 - in Cohort 2 2+1 Schedule subjects
Respiratory tract infection (Infections and infestations) | 5 | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Unsolicited AE reported during the 31-day post-vaccination period in Cohort 1
Conjunctivitis (Infections and infestations) | 0/0 | 0/0 | 6 | 4 | 10 | 6 | 0/0 | 0/0 — Unsolicited AE reported during the 31-day post-vaccination periods, across doses - in Cohort 2 3+0 Schedule subjects
Respiratory tract infection (Infections and infestations) | 0/0 | 0/0 | 80 | 68 | 80 | 80 | 0/0 | 0/0 — Unsolicited AE reported during the 31-day post-vaccination periods, across doses - in Cohort 2 3+0 Schedule subjects
Upper respiratory tract infection (Infections and infestations) | 0/0 | 0/0 | 12 | 14 | 12 | 10 | 0/0 | 0/0 — Unsolicited AE reported during the 31-day post-vaccination periods, across doses - in Cohort 2 3+0 Schedule subjects
Respiratory tract infection (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 56 | 58 — Unsolicited AE reported during the 31-day period after vaccination with the first 2 doses - in Cohort 2 2+1 Schedule subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.